## Statistical Analysis Plan

Protocol Number: MT-5547-J01

A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain

For database at week 16

Version: 2.0

Date: 2 July 2020

For database at week 68

Version: 1.0

Date: 19 April 2021

NCT number: NCT03245008

## Statistical Analysis Plan (For Database at Week 16)

## List of Errata

Protocol No. MT-5547-J01

A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain

| Prepared By: | Mitsubishi Tanabe Pharma Corporation |
|--------------|--------------------------------------|
| Version: | 2.0 |
| Date: | 2-July-2020 |

NCT Number: NCT03245008

## APPROVAL FORM

## Statistical Analysis Plan(For Database at Week 16)

## -List of Errata-

|---|---|
| Protocol Title | A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain |
| Version / Date | 2.0 / 2-July-2020 |

## Authors:

| Statistics Author | |
|-------------------|-----------------|
| Print Name: | |
| Position: | Biostatistician |

#### Approved by:

| Responsible Biostatistician |
|-----------------------------|
| Refer to email |
| Refer to email |

## 1. INTRODUCTION

This list of errata is based on the statistical analysis plan for database at week 16 dated 10-February-2020.

## 2. LIST OF ERRATA

| befroe change | after change |
|---|---|
| 8.2.1. Primary Efficacy Endpoint | 8.2.1. Primary Efficacy Endpoint |
| Sensitivity analyses | Sensitivity analyses |
| <ul> <li>Multiple Imputation (MI) analysis by</li> </ul> | Multiple Imputation (MI) analysis by |
| Reason for Discontinued Treatment | Reason for Discontinued Treatment |
| The following SAS code will be used to | The following SAS code will be used to |
| generate the monotone missing data pattern: | generate the monotone missing data pattern: |
| 10. CHANGE FROM THE PROTOCOL | 10. CHANGE FROM THE PROTOCOL |
| | Sensitivity analysis of the primary endpoint |
| There are currently no changes to analysis | was changed from placebo multiple |
| from protocol. | imputation analysis to multiple imputation |
| | analysis with values centered at the mean |
| | baseline value of the treatment group by |
| | reason for discontinued treatment. Because |
| | confirming the robustness against missing |
| | data using the multiple imputation method |
| | similar to the primary analysis in the overseas |
| | P3 study. |

#### 3. HISTORY OF ERRATA

## <u>Up to version 1.0 (24-April -2020)</u>

| befroe change | after change |
|---|---|
| 4.2. Final Analysis | 4.2. Final Analysis |
| This SAP for 16 week will be finalized | This SAP for 16 week will be finalized before |
| before database lock in week 16. The | database lock in week 16. The efficacy |
| efficacy analysis performed at week 16 is the | analysis performed at week 16 is the final |
| final efficacy analyasis. | efficacy analysis. |
| 7.1.1.1. Demographic and Other Baseline | 7.1.1.1 Demographic and Other Baseline |
| Characteristics | Characteristics |
| (3)Time since osteoarthritis diagnosis (years) | (3) Time since osteoarthritis diagnosis (years) |
| If (month of date of consent > month of | If (month of date of consent > month of |
| osteoarthritis diagnosis) or (month of date of | osteoarthritis diagnosis) or (month of date of |
| consent = month of date osteoarthritis | consent = month of date osteoarthritis |
| diagnosis, and day of date of consent >= day | diagnosis, and day of date of consent >= day |
| of date of osteoarthritis diagnosis), then | of date of osteoarthritis diagnosis), then Time |
| Time since osteoarthritis diagnosis (years) = | since osteoarthritis diagnosis (years) = <del>year of</del> |
| year of date of consent – year of date of | (date of consent – <del>year of</del> date of osteoarthritis |
| osteoarthritis diagnosis | diagnosis <u>)/365.25*</u> |
| if else case, then Time since osteoarthritis | if else case, then Time since osteoarthritis |
| diagnosis (years) = year of date of consent - | diagnosis (years) = <del>year of (</del> date of consent – |
| year of date osteoarthritis diagnosis – 1. | <del>year of</del> date osteoarthritis diagnosis – 1) |
| | <u>/365.25*</u> . |
| | * 1 year = 365.25 days |
| 7.1.1.2. Treatment Duration and Compliance | 7.1.1.2. Treatment Duration and Compliance |
| 1)Treatment Duration (days) = The date of | 1)Treatment Duration (days) = The date of last |
| last study drug injection prior to week 16 - | study drug injection prior to week 16 - the |
| the date of the first study drug injection + | date of the first study drug injection + min(28 |
| min(28 or (the date of last study drug | or (the date of week 16 study drug infection - |
| infection - the date of Week 16 study drug | the date of <u>last</u> study drug injection <u>prior to</u> |
| injection)) | week 16)) |
| 7.1.2.6. SF-36 / EQ-5D-5L | 7.1.2.6. SF-36 / EQ-5D-5L |
| e.g ) If answer is [1 1 1 1 1], Utility Index | e.g ) If answer is [1 1 1 1 1], Utility Index |
| Score is=1+0+0=1. If answer is [1 1 3 2 1], | Score is=1+0+0=1. If answer is [1 1 3 2 1], |

| Utility Index Score | Utility Index Score |
|---|---|
| is=1+(-0.060924)+(-0.091131-0.068178)=0. | is=1+(-0.060924)+(-0.091131-0.0 <u>44545</u> )=0. <u>8</u> |
| 779767. | <u>034</u> . |
| 8.1.4. Treatment Duration and Compliance | 8.1.4. Treatment Duration and Compliance |
| Treatment compliance will be summarized | Treatment compliance will be summarized by |
| by treatment group and combined MT-5547 | treatment group and combined MT-5547 on |
| on the SAF population. | the <u>FAS</u> population. |

#### APPROVAL FORM

#### Statistical Analysis Plan(For Database at Week 16)

#### -List of Errata-

|---|---|
| Protocol Title | A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain |
| Version / Date | 2.0 / 2-July-2020 |

#### Authors:

| Statistics Author | |
|-------------------|-----------------|
| Print Name: | |
| Position: | Biostatistician |

#### Approved by:

| Statistic Approver | |
|--------------------|-----------------------------|
| Print Name: | |
| Position: | Responsible Biostatistician |
| Signature: | Refer to email |
| Approval date: | Refer to email |

# Statistical Analysis Plan (For Database at Week 16)


A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain

| Prepared By: | Mitsubishi Tanabe Pharma Corporation |
|--------------|--------------------------------------|
| Version: | 1.0 |
| Date: | 10-February-2020 |

## APPROVAL FORM

## Statistical Analysis Plan

|---|---|
| Protocol Title | A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain |
| Version / Date | 1.0 / 10-February -2020 |

#### Authors:

| Statistics Author | | · |
|-------------------|-----------------|---|
| Print Name: | | |
| Position: | Biostatistician | |

Approved by:

| Approved by. | |
|--------------------|-----------------------------|
| Statistic Approver | |
| Print Name: | |
| Position: | Responsible Biostatistician |
| Signature: | |
| Approval date: | |

## TABLE OF CONTENTS

| 1. | INTRODUCTION | 7 |
|---|---|---|
| 2. | STUDY OBJECTIVE AND ENDPOINTS | 7 |
| | 2.1. Study Objective(s) | 7 |
| | 2.2. Study Endopoint(s) | 7 |
| | 2.2.1. Efficacy Endpoint(s) | 7 |
| | 2.2.2. Safety Endpoint(s) | 8 |
| 3. | STUDY DESIGN | 8 |
| | 3.1. Study Design | 8 |
| | 3.2 Schedule of Study Procedures | 9 |
| | 3.2.1. Test/Observation Schedule | 9 |
| | 3.3. Sample Size and Power Considerations | 14 |
| 4. | PLANNED ANALYSIS | 17 |
| | | 17 |
| | 4.1. Interim Analysis | 1 /<br>1 <b>7</b> |
| | 4.2. Final Analysis | 1 /<br>1 <b>7</b> |
| | 4.3. Independent Data Monitoring Board | 1 / |
| 5. | ANALYSIS POPULATIONS | 17 |
| 6. | STATISTICAL CONSIDERATIONS | 19 |
| | 6.1. Descriptive Statistics | 19 |
| | 6.2. Statistical Tests | 19 |
| 7. | DATA CONVENTIONS | 19 |
| | 7.1. Analysis Variable Definitions | 19 |
| | 7.1.1. Study Subjects | 19 |
| | 7.1.1. Study Subjects | 19 |
| | 7.1.1.2. Treatment Duration and Compliance | 20 |
| | 7.1.2. Efficacy assessments | 20 |
| | 7.1.2.1. WOMAC pain subscale score | 20 |
| | 7.1.2.1. WOMAC pain subscale score | 20 |
| | 7.1.2.3. WOMAC physical function subscale score | 20 |
| | 7.1.2.4. WOMAC stimess subscale score | 20 |
| | 7.1.2.5. NRS score 21 | |
| | 7.1.2.6. SF-36 / EQ-5D-5L | 2.1 |
| | 7.1.2.7. Response rate based on the OMERACT-OARSI criteria | 23 |
| | 7.1.2.8. Rescue Medication | 23 |
| | 7.1.2.3. Rescue Medication | 23 |
| | 7.1.3.1. Adverse Events | 22 |
| | 7.2. Analysis Visit Definitions | 24 |
| | 7.2. Analysis visit Definitions 7.3. Data Handling Convention for Missing Data | 25 |
| | 7.3. Data Handing Convention for missing Data | |

| 8.1. Study Subjects | |
|---|---|
| <ul><li>8.1.1. Subject Disposition</li><li>8.1.2. Analysis Populations</li><li>8.1.3. Demographic and Other Baseline Characteristics</li></ul> | |
| 8.1.2. Analysis Populations | |
| 8.1.3. Demographic and Other Baseline Characteristics | 25<br>27<br>27 |
| 8 1 4. Treatment Duration and Compliance | 27<br>27<br>27 |
| | 27<br>27 |
| 8.2. Efficacy Assessments | 27 |
| 8.2.1. Primary Efficacy Endpoint | 34 |
| 8.2.2. Key Secondary Efficacy Endpoints | |
| 8.2.3. Other Efficacy Endpoints | 34 |
| 8.3. Safety Assessments | 36 |
| 8.3.1. Adverse Events | 36 |
| 9. DATA PRESENTATION CONVENTIONS | 37 |
| 9.1. Number of Digits to Report | 37 |
| 9.2. Treatments to Report | 37 |
| 9.3. Analysis Visits to Report | 37 |
| 10. CHANGE FROM THE PROTOCOL | 38 |
| 11. SOFTWARE | 38 |
| 12. REFERENCES | 38 |
| 13. APPENDIX | 39 |
| 13.1. SF-36v2 Scoring Algorithm <sup>[2]</sup> | 39 |

## **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|-----------------------------------------------------|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine transaminase |
| ALP | Alkaline phosphatase |
| ANCOVA | Analysis of covariance |
| AST | Aspartate transaminase |
| ATC | Anatomical therapeutic chemical |
| BDR | Blinded data review |
| BLQ | Below limit of quantification |
| BMI | Body mass index |
| CI | Confidence interval |
| DA | Destructive arthropathy |
| DP | Decimal places |
| DMC | Data monitoring committee |
| EQ-5D-5L | EuroQol Group Questionnaire |
| FAS | Full analysis set |
| ITT | Intent-to-treat |
| K-L | Kellgren-Lawrence |
| LLOQ | Lower limit of quantitation |
| MAR | Missing at random |
| MedDRA | Medical dictionary for regulatory activities |
| MMRM | Mixed model repeated measures |
| NGF | Nerve growth factor |
| NRS | Numerical rating scale |
| NSAID | Nonsteroidal anti-inflammatory drug |
| OMERACT-OARSI | Outcome Measures in Rheumatology Arthritis Clinical |
| | Trials-Osteoarthritis Reseach Society International |
| PGA | Patient Global Assessment |
| PPS | Per protocol set |
| PT | Preferred term |
| q4w | Every 4 weeks |
| q8w | Every 8 weeks |
| QOL | Quality of life |
| RAND | All subjects randomized population |
| RPOA | Rapidly progressive osteoarthritis |
| SAE | Serious adverse event |
| SAF | Safety population |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SF-36 | Short form 36-item health survey |
| SIF | Subchondral insufficiency fracture |
| SOC | System organ class |

| TESAE | Treatment emergent serious adverse events |
|-------|----------------------------------------------------------------|
| ULN | Upper limit of normal range |
| WHO | World Health Organization |
| WOMAC | Western Ontario and McMaster Universities Osteoarthritis Index |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol (v4.0) dated 31-July-2018. This protocol will plan to respectively perform the statistical analysis for the clinical trial data from screening to Week 16, from screening to Week 24 and from screening to Week 48.

For the clinical trial data from screening to Week 16, this SAP covers statistical analysis, tabulations of the study data to investigate the efficacy and safety of MT-5547 SC 1mg q4w and 1mg q8w compared to matching placebo. Therefore, this SAP will be finalized prior to database lock at Week16 to ensure the credibility of the study results by pre-specifying the statistical methods for the data analyses before un-blinding of treatment assignments. For the clinical trial data from screening to Week 24 and from screening to post-treatment observation period of Week 20 after the end of the treatment period, the other SAPs will be separately created.

Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

#### 2. STUDY OBJECTIVE AND ENDPOINTS

#### 2.1. Study Objective(s)

The objective of this study is to verify the superiority of 16 weeks of MT-5547 treatment to placebo, as evidenced by the WOMAC pain subscale score (the efficacy outcome measure), in patients with osteoarthritis of the knee or hip. Additional objectives of the study are to investigate the efficacy, safety, and pharmacokinetics of MT-5547 in long-term use.

#### 2.2. Study Endopoint(s)

#### 2.2.1. Efficacy Endpoint(s)

- (1) Primary efficacy endpoint
  WOMAC pain subscale score (change from baseline at Week 16)
- (2) Key secondary efficacy endpoint WOMAC physical function subscale score (change from baseline at Week 16)
- (3) Secondary efficacy endpoints
  - 1) Patient global assessment (PGA) (change from baseline at each assessment time point)
  - 2) WOMAC pain subscale score (change from baseline at each assessment time point)
  - 3) WOMAC physical function subscale score (change from baseline at each assessment time point)
  - 4) WOMAC stiffness subscale score (change from baseline at each assessment time point)
  - 5) WOMAC total score (change from baseline at each assessment time point)
  - 6) Proportions of subjects with 30%, 50%, 70% and 90% improvements in their WOMAC pain subscale scores compared to baseline (Weeks 16)
  - 7) Proportions of subjects with 30%, 50%, 70% and 90% improvements in their WOMAC physical function subscale scores compared to baseline (Weeks 16)

- 8) Numerical Rating Scale (NRS) score for the mean pain on walking in the evaluated joint (change from baseline at each assessment time point)
- 9) SF-36 (change from baseline at each assessment time point)
- 10) EQ-5D-5L (change from baseline at each assessment time point)
- 11) Improvement rate based on the Outcome Measures in Rheumatology Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) criteria (at Weeks 16)
- 12) Amount of rescue medication used (number of days on which rescue medication was used, and amount [number of tablets] used)

#### 2.2.2. Safety Endpoint(s)

- (1) Adverse events and adverse reactions
- (2) Adverse events of special interest as defined in the protocol i.e. adjudicated arthropathy, sympathetic nervous system disorders and altered peripheral sensation.

#### 3. STUDY DESIGN

#### 3.1. Study Design

Study Phase: Phase 2/3

Type of Study: Confirmatory Study

Parallel group, randomized, placebo-controlled, double-blind (24 weeks), multicenter





- 1) The post-treatment observation period will be the 20 weeks from the day after the end of the 48-week treatment period. Furthermore, for subjects discontinued from the study, the post-treatment observation period will be the 24 weeks from the administration of MT-5547 or MT-5547 placebo. If a joint replacement procedure is going to be performed, the postoperative test observation period will be the period from the day after the day of discontinuation until 20 weeks after the joint replacement procedure is performed.
- 2) From Week 16 to Week 48, the placebo group will receive an additional dose of naproxen tablets to reduce the dropout rate in the placebo group. The MT-5547 group will receive an additional dose of naproxen placebo tablets.

For each subject, the data for up through Week 16 will be fixed prior to the Week 20 visit, and the fixed data will be prepared.

3) The blind will be maintained, including for the study sponsor, until the key code is opened after the data have been fixed for all subjects in Week 24. In addition, in order to eliminate any bias that could affect the study assessments, to the extent possible, the blind will be maintained with respect to the study site and the subject even after the opening of the study sponsor key code.

#### 3.2. Schedule of Study Procedures

#### 3.2.1. Test/Observation Schedule

Statistical Analysis Plan Protocol No. MT-5547-J01

Mitsubishi Tanabe Pharma Corporation (1) Test/Observation Schedule from informed consent to Week 48 of treatment period (if a joint replacement procedure is not going to be performed)

| | | | | | | | Tenator | Transferent negation | ١ | | | - | | | | Treatment period | period | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Inform | Screening | Pre-treatment<br>of observation | Day1 | Week1 | Week2 | Week4 | _ | Week12 | Week16 | Week 20 | Week 24 | Week 28 | Week 32 | Week 36 | Week 40 Week 44 | Week 44 | Week 48 | At<br>withdrawa |
| | P | | period | Baseline | | | - | - | _ | - | - | 1 | 1 | 1 | 1 | į | 92. | 11.00 | <u>*</u> _ |
| Visit times (visit window) | + | Day -37<br>~ -8 | Day -7 ~~-1<br>(±3) | | E gá | Day 15<br>(43) | Day 29<br>(±7) | Day 57<br>(±7) | Day85<br>(#7) | Day 113<br>(#7) | Day 141<br>(#7) | Day 169 | Day 197<br>(±7) | Day 225<br>(#7) | Day 253<br>(±7) | (#1) | (#) | (#1) | |
| Visit Number | | - | 7 | 3 | 7 | s | 9 | 7 | | • | 2 | = | 12 | 22 | 7 | 22 | 16 | 17 | |
| Written informed consent | × | | | | | | 1 | | 1 | 1 | T | | T | | | | | | |
| Eligibility confirmed | 1 | × | × | ×, | | Ī | T | | 1 | İ | T | T | Ī | Ī | Ī | | | | |
| Demographics | I | × | | × | | T | t | T | | T | Ī | | | Ī | | | | | |
| Randomization | İ | | | < × | | 1 | × | × | × | × | × | × | × | × | × | × | x | | |
| Study drug SC administration | I | | | | | | | | | V | | | | | | | | Î | |
| Administration of naproxen | İ | | | | | | T | | | × | × | × | × | × | × | × | x | | |
| Detroit of naproxen | | | | | | | | | | | × | × | × | × | × | × | × | х | × |
| Delivery of acetaminonhen | | | × | × | | × | × | × | × | × | × | × | × | х | x | × | х | | |
| Return of acetaminophen/check of | | | | × | | × | × | × | × | × | × | × | × | × | х | × | × | × | × |
| amount taken | | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| [Rifferey] | | | | | | 1 | | | | | | | | | | | | | |
| MDS (exercise della main) | | | × | Ŭ. | | T | | | ľ | 1 | | | | | | | | | |
| WOMAC | | × | | x | × | × | х | × | × | × | × | × | × | × | × | × | × | × | × |
| PGA of OA | | х | | X | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| SF-36 | | | | × | | | × | × | | × | | × | | × | | × | | × ; | < |
| EQ-5D-SL | | | | × | | | × | × | | × | | Ĭ | 1 | × | 1 | ¥ | | 4 | 4 |
| [Safety] | | | | | | Ī | | | ľ | | | 1 | | ſ | | | | | |
| Body weight (height: only at screening) | _ | × | | | | | | | | × | | | | | | | | × | × |
| Vital day | | × | | × | × | × | × | × | × | × | × | х | х | × | x | × | × | × | × |
| RCG | | × | | | | | | | | | | | | | | | | × | × |
| Physical examination | | × | | | | | | | | | | × | | × | | | | × | × |
| Orthostatic blood pressure | | × | х | × | | x | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Injection site assessment | | | | × | | | × | × | × | × | × | х | Х | X | × | × | × | | |
| Joint Pain Questionnaire | | × | | × | × | x | x | x | × | × | × | × | x | × | × | × | × | × | × |
| Autonomic Nerve Ouestionnaire | | × | | × | | | × | × | x | x | x | × | × | × | × | × | × | × | × |
| Neurological evaluation | | × | i | X<br>(brief | | X<br>(brief | X<br>(brief | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | X<br>(brief<br>version) | × | × |
| Radiology (bilateral knees, hips, | | × | | | | | | | - | × | | | | | | | | x | х |
| shoulders)'<br>MRI testing | | | | | | | | | | | | | | | | | | | |
| (evaluated joint, contralateral joint, | | × | | | | | | | | | | | | | | | | | |
| MRI testing (joint of joint replacement | = | | | | | | | | | | | | | | | | | | × |
| Adverse events | Ĺ | | | | | | | | | | | | | | | | | $\uparrow$ | × |
| At joint pain wersoning | | | | | \<br>↓ | | | | | | | | | | | | | $\uparrow$ | × |
| (finaging [X-ray, MRI] assessments) | | | | | | | | | | | | | | | | | | | × |
| Laboratory testing | | × | | × | | | × | × | × | × | | × | Ì | × | | × | | × | × |
| Pregnancy test (for WOCBP)11 | | × | | х | | | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Bone density <sup>12</sup> | | × | | | | | | | | | | | | | | | | × ; | × : |
| Urinalysis | | × | | × | | | | | | × | | × | | | | | | × | × |
| [Pharmacokinetics] | | | | | | | - | | | ; | | 2 | | 1 | | 1 | SP. | , | , |
| PK measurements | $\int$ | | | X | × | × | χ | × | × | × | | X | | Ł | | × | × | 4 > | < × |
| ADA antibody | _ | | | ķ | | | | | | × | | × | | | | | | 4 | • |
| [Other] | | | | | | | | | | | | | | | | | | | ¥ |
| | - | | | - | | | 1 | | | - | | <br> | | <u> </u> | | | | | 1 |
| | 4 | | | - | | | | | | | | | | | | | | | |

Page 10 of 43

(2) Test/Observation Schedule of post-treatment observation period (if a joint replacement procedure is not going to be performed)

| | Po | st-treatmen | t observati | on period ( | 20 weeks)14 | |
|---|---|---|---|---|---|---|
| | Week 52 | Week 56 | Week 60 | Week 64 | Week 68 | At<br>withdra<br>wal |
| Visit times (visit window) | Day 365<br>(±7) | Day 393<br>(±7) | Day 421<br>(±7) | Day 449<br>(±7) | Day 477<br>(±7) | |
| Visit Number | 18 | 19 | 20 | 21 | 22 | |
| Written informed consent | | | | | | |
| Eligibility confirmed | | | | | | |
| Demographics | | | | | | |
| Rando mization 1 | | | | | | |
| Study drug SC administration <sup>2</sup> | | | | | | |
| Administration of naproxen | | | | | | |
| Delivery of naproxen | | | | | | |
| Return of naproxen | | | | | | |
| Delivery of acetaminophen | | | | | | |
| Return of acetaminophen/check of | | | | | ] | |
| amount taken <sup>3</sup> | | | | | | |
| Concomitant medications | X | X | X | X | X | X |
| [Efficacy] | | | | | | |
| NRS (average daily pain)4 | | | | | | |
| WOMAC <sup>5</sup> | X | | X | | X | X |
| PGA of OA | X | | X | | X. | X |
| SF-36 | | | | | X | X |
| EQ-5D-5L | | | | | X | X |
| [Safety] | | | | | | |
| Body weight (height: only at screening) | | | | | x | X |
| Vital signs <sup>6</sup> | X | | | | X | X |
| ECG | | | | | | |
| Physical examination | _ | | | | X | X |
| Orthostatic blood pressure | X | | | | X | X |
| Injection site assessment | | | | | | i |
| (30 minutes after administration) | | | | | | |
| Joint Pain Questionnaire | X | ļ | | | X | X |
| Autonomic Nerve Questionnaire | X | | <u> </u> | ļ | X | X |
| Neurological evaluation | X<br>(brief<br>version) | | | | x | x |
| Radiology (bilateral knees, hips, | | | | | x | x |
| shoulders) <sup>7</sup> MRI testing | | | _ | | ^ | A |
| (evaluated joint, contralateral joint, knee or hip joints with K-L ≥ 3) <sup>7</sup> | 1 | | | | 1 | |
| MRI testing (joint of joint replacement | | | | | | x |
| Adverse events | ← | 1 | | 1 | $\rightarrow$ | X |
| At joint pain worsening | | 1 | <b>T</b> | | | |
| (imaging [X-ray, MRI] assessments)8 | <del></del> | | | | <del> </del> | X |
| JOA Score | | | | | | X |
| Laboratory testing 10 | T - | | | | X | X |
| Pregnancy test (for WOCBP) <sup>11</sup> | x | 1 | | | X | X |
| Bone density 12 | | | | | | |
| Urinalysis | <del> </del> | 1 - | <u> </u> | † - | x | X |
| [Pharmacokinetics] | t | | | | | |
| PK measurements | x | X | 1 | Ι | X | X |
| | | <del> </del> | <u> </u> | | X | X |
| ADA antibody [Other] | <del> </del> | <del></del> | <u> </u> | | 1 23 | |
| [Omer] | <del> </del> | т — | | 1 | T <b>m</b> | 1 = |

- 1) Subjects will be randomized (enrolled at the start of the treatment period) after all of the assessments through the pre-treatment observation period have been completed.
- 2) Investigational drug or comparative drug will be administered subcutaneously after all of the safety assessments, efficacy assessments, and collection of blood samples for pharmacokinetic assessments have been completed, and subjects will be kept under supervision at the study site for 30 minutes after the administration of the study drug.
- 3) The dose of acetaminophen taken will be checked based on the treatment diary. Every night, subjects will record in their treatment diaries the amount (number of tablets) of acetaminophen they took that day.
- 4) Every night (and as a rule at the same time) from the start of the pre-treatment observation period until Week 16, subjects will use the IVRS to report the mean pain on walking for the previous 24 hours (NRS data). Subjects will receive instruction in how to use the IVRS on the day of the visit at the start of the pre-treatment observation period.
- 5) The WOMAC score at screening will be assessed for the right knee joint, the left knee joint, the right hip joint, and the left hip joint, and the evaluated joint will be determined based on the WOMAC pain subscale scores. At the other time points, the WOMAC score will be assessed for the evaluated joint only.
- 6) If the pulse is less than 45 bpm at an assessment time point after investigational drug or comparative drug administration, electrocardiography will be performed and the patient carefully examined for cardiac function abnormalities.
- 7) Screening:

The following imaging tests will be performed for subjects who meet the study eligibility criteria, and the images will be submitted to a central laboratory. Imaging tests will also be performed if the central laboratory requests that additional tests be conducted.

- · X- ray tests: Both knee joints, both hip joints, both shoulder joints
- MRI tests: The evaluated joint, the joint opposite the evaluated joint, and any knee or hip joints with a K-L grade of 3 or more

MRI tests will be performed as needed by the (sub)investigator.

A check will be performed by the day specified below to make sure that the results of the central assessments meet the study enrollment criteria.

- · X-ray tests: By the start of the pre-treatment observation period
- · MRI tests: By baseline

If the results of the central assessments cannot be confirmed by the specified day, then re-screening will be performed.

#### Baseline and after baseline:

At week 16, 48 (or at the early termination of the treatment period) and at 68 weeks (or at the early termination of the post-treatment observation period), images will be submitted to the central laboratory. If the (sub)investigator determine that there is an abnormal finding compared to normal osteoarthritis, MRI tests will be performed as needed. The images will be submitted to a central laboratory. Imaging tests will also be performed if the central laboratory requests that additional tests be conducted, and the images submitted to the central laboratory(for more detailed information, see in the text "9.2.4.1.11 Imaging Tests").

#### Week 16:

The X-ray tests (both knee joints, both hip joints, both shoulder joints) will be performed by the (sub)investigator. The (sub)investigator will check the X-ray images before administered the investigational drug or comparative drug to determine whether or not investigational drug or comparative drug should be administered. If any abnormalities are found, investigational drug or comparative drug administration will be postponed. If the central laboratory rules out adjudicated arthropathy, investigational drug or comparative drug administration will be resumed.

Assessment at the early termination of the treatment period and the early termination of the post-treatment observation period

The X-ray tests (both knee joints, both hip joints, both shoulder joints) will be performed by the (sub)investigator. The images will be submitted to a central laboratory. If more than 30 days have passed since the last images were taken, images will be taken again. If not more than 30 days have passed, imaging tests will be performed if the (sub)investigator determines that it is necessary.

13)

If joint replacement surgery is required, the MRI tests of the joint of surgery will be performed (for more detailed information, see in the text "9.2.4.1.13 Assessments if a Joint Replacement Procedure Is Scheduled").

- 8) If a subject experiences a sudden worsening of pain that would not occur in the normal course of osteoarthritis, the (sub)investigator will postpone investigational drug or comparative drug administration, and perform imaging test (X-ray and MRI) of the affected joint. Imaging test (X-ray and MRI) of other joints will be performed as needed by the (sub)investigator. Imaging tests will also be performed if the central laboratory requests that additional tests be conducted. All images will be submitted to the central laboratory. The results of the central assessment will be checked by the (sub)investigator. The investigational drug or comparative drug administration will be postponed until the central laboratory rules out adjudicated arthropathy. If the result of the central assessment is adjudicated arthropathy, then study treatment must be discontinued. If adjudicated arthropathy is ruled out by the central assessment, the (sub)investigator will determine whether or not study treatment should be continued.
- Assessmets of the joint by JOA score at discontinuation will be performed for subjects who required joint replacement surgery during the study.
- 10) Hematology and blood biochemistry tests will be performed. HbA1c, HBs antigen, HBs antibody, HCV antibody, and HIV antibody will be measured only at screening.
- 11) At screening, the pregnancy test will be performed using serum. At all other time points, the pregnancy test will be performed using urine. Furthermore, pregnancy tests will not be performed for postmenopausal females who have been amenorrheic for at least 1 year or for females who have undergone a surgical hysterectomy or bilateral ovariectomy. If a positive result is obtained on a urine pregnancy test, a serum pregnancy test will be performed. If a negative result is obtained on a serum pregnancy test, the study can be continued for the patient. If the serum pregnancy test is also positive, study treatment will be discontinued.
- 12) Bone density will be measured only at those study sites that are capable of performing measurements using the DEXA method. If it can not be measured at screening priod, it may be measured during the pre-treatment observation period.

14) The Week 64 assessments may be performed by telephone.

- 15) The blood samples will be collected before the investigational drug or comparative drug is administered.
- 16) In the case of early termination of the treatment period, follow-up evaluation of the same item as at the time of visit of the corresponding completed subjects below is carried out 4, 8, 12, 16, 20 and 24 weeks after the last dose of the investigational drug or comparative drug. However, blood sample collection for pharmacokinetic evaluation is performed only 24 weeks after the last dose (blood sample collection for PK measurement is not necessary 4, 8 and 12 weeks after the the last dose corresponding to treatment period 48, 52 and 56 weeks of the completed subjects). The visit window at each evaluation time point is plus or minus 7 days.

| Early termination of the treatment period | 4 weeks<br>after the<br>last dose | 8 weeks<br>after the<br>last dose | 12 weeks<br>after the<br>last dose | 16 weeks<br>after the<br>last dose | 20 weeks<br>after the<br>last dose | 24 weeks<br>after the<br>last dose | the early<br>termination of the<br>post-treatment<br>observation period |
|---|---|---|---|---|---|---|---|
| Completed of the treatment period | Week 48 | Week 52 | Week 56 | Week 60 | Week 64 | Week 68 | the early<br>termination of the<br>post-treatment<br>observation period |

When assessments at discontinuation is included in visit window of each assessment time point, the same ones as those normally assessed at discontinuation. After assessment at discontinuation, the same ones as those normally assessed at the last dose of investigational drug or comparative drug.

If more than 30 days have passed since the last images were taken, images will be taken again. If not more than 30 days have passed, imaging tests will be performed if the (sub)investigator determines that it is necessary.

The tests at discontinuation and post-joint replacement procedure test/observation will be performed for

- subjects who required joint replacement surgery during the study. The all images will be submitted to a central laboratory (for more detailed information, see "10 (3) Post-joint replacement procedure test/observation schedule). If the assessments at discontinuation are not performed before the joint replacement procedure is performed, then images from before the procedure will be obtained and sent to the central laboratory.
- 17) The screening period is from "the screening start date" to the day before "the pre-treatment of observation period start date", and the screening start date and the end date are defined along with the allowable range of "the pre-treatment of observation period" (for example, when the pre-treatment of observation period is 4 days, The maximum screening period is 30 days from Day 34 to Day 5, the pre-treatment of observation period is 10 days, the screening period is the maximum from Day 40 to Day 11).

At each study visit after the baseline date, the assessments that are performed by the subjects themselves (WOMAC, PGA, joint pain survey, SF-36, EQ-5D-5L, survey of autonomic symptoms) will be performed before all of the other assessments (including the assessments that are performed by the (sub)investigator) (except for cases where imaging tests are performed on a different day).

#### (3) Post-joint replacement procedure test/observation schedule

| | After surgery <sup>1</sup> | Long-term <sup>1</sup> |
|---|---|---|
| Follow-up day (visit window) | Follow-up survey, 4 weeks post-<br>operative | Follow-up survey 2, 20 weeks post-<br>operative |
| · . | 29 days post-operative (±5 days) | 141 days post-operative (±7 days) |
| Concomitant medications | X | X |
| [Safety] | | |
| Vital signs | X | X |
| Joint Pain Ouestionnaire | X | X |
| JOA score <sup>2</sup> | x | X |
| Radiology (bilateral knees, hips, shoulders) | X | X |
| Adverse events | <del></del> | $\rightarrow$ |
| At joint pain worsening (imaging [X-ray, MRI] assessments)3 | <del>-</del> | <b>──</b> |

- 1) Information about the procedure, including prosthesis replacement and/or the extent of surgery wound healing, will be collected.
- 2) The condition of the joint following joint replacement surgery will be assessed using the JOAScore.
- 3) If a sudden worsening of pain that does not occur in the normal progression of osteoarthritis occurs, the (sub)investigator will perform imaging test (X-ray and MRI) of the affected joint. Imaging test (X-ray and MRI) of other joints will be performed as needed by the (sub)investigator. Imaging tests will also be performed if the central laboratory requests that additional tests be conducted. All images will be submitted to the central laboratory.

#### 3.3. Sample Size and Power Considerations

The original target sample size is 568 treated subjects (142 subjects per group)
(MT-5547 1 mg q4w group: 142 subjects; MT-5547 3 mg q4w group: 142 subjects;
MT-5547 6 mg q8w group: 142 subjects; placebo group: 142 subjects)

After initiation of this study, based on the recommendations from the IDMC, the 3 mg q4w and 6 mg q8w groups were removed and 1 mg q8w group was newly added to the treatment

groups.

The amended target sample size is 506 treated subjects, including the subjects who were randomized to 1 mg q4w/placebo groups before the amendment (approximately 40 subjects per group) and the subjects who are randomized to 1 mg q4w/1 mg q8w/placebo groups with the ratio of 1:1:1 after the amendment (142 subjects per group).

(MT-5547 1 mg q4w group: 182 subjects; MT-5547 1 mg q8w group: 142 subjects; placebo group: 182 subjects)

In addition, 57 patients each were enrolled in the MT-5547 3 mg q4w and 6 mg q8w groups prior to the protocol amendment (Ver. 04.00.00000) and were discontinued from study drug based on the recommendations from the IDMC. Thus, enrollment of 563 subjects is planned for this study in total.

#### The original rationale at the initiation of the study

Because this study is being conducted as a placebo-controlled study, in order to detect a statistical difference between the MT-5547 groups and the placebo group, the mean intergroup difference relative to placebo in both the change from baseline in the WOMAC pain subscale score and the change from baseline in the physical function subscale score at Week 16 for the MT-5547 3 mg SC q4w, 6 mg SC q8w, and 1 mg SC q4w groups was set at 1.1, and the standard deviation 2.5, on the basis of the results obtained in the overseas P2a study (R475-PN-0901) and the overseas P2b study (R475-PN-1227) (Table 3.3-1). The effect relative to placebo in the P3 study of 5 mg and 10 mg of tanezumab, another NGF inhibitor, was 0.81 to 1.21 in the WOMAC pain subscale score and 0.98 to 1.25 24), 25) in the WOMAC physical function subscale score, and it therefore appears that a mean difference between the MT-5547 groups and placebo of 1.1 is a realistic assumption. It also appears that the minimum clinically significant difference in each WOMAC score will be around 0.67 to 0.75 <sup>26), 27)</sup>. The aforementioned intergroup difference of 1.1 exceeds the minimum clinically significant difference, and therefore seems to be an appropriate value to use for the intergroup difference. Based on a one-sided significance level of 2.5% and multiplicity adjustment based on a gate keeping method using a graphical approach, the power for MT-5547 3 mg SC q4w, 6 mg SC q8w, and 1 mg SC q4w will be 90%, 88%, and 88%, respectively, for the primary endpoint, and 82%, 79%, and 79%, respectively, for the key secondary endpoint. A 2-sample t-test will be used for the tests in each step. Based on this assumption, the number of subjects who will complete 16 weeks of treatment in each group will be 120.

Furthermore, because the proportion of missing data for the primary endpoint and the key secondary endpoint at Week 16 is around 15% according to Table 3.3-1, it is being assumed that the proportion of missing data at Week 16 will be 15%, and the number of patients per

group is therefore being set at 142.

#### The rationale after the changes in treartment groups

Assuming the absolute treatment difference of 1.1 between the MT-5547 1 mg SC q8w groups and placebo in both the change from baseline in the WOMAC pain subscale score and the change from baseline in the physical function subscale score at Week 16 with an associated standard deviation of 2.5 based on the original rationale at the initiation of the study, the number of patients per group after the protocol amendment (Ver. 04.00.00000) is planned to 142 subjects per group. The structure of statistical hypotheses have been changed due to the removal of 3 mg q4w / 6 mg q8w groups and the addition of 1 mg q8w. It is noted that approximately 40 subjects per group were randomized to 1 mg q4w / placebo groups before the amendment. For evaluation on 1 mg q4w, since subjects are randomized to 1 mg q4w / placebo at the same time with the same ratio of 1:1 regardless of pre- or postamendment, analyses will be performed with pooled comparable data including pre- and postamendment data on 1 mg q4w / placebo (1 mg q4w group: 182 subjects; placebo group: 182 subjects). For evaluation on 1 mg q8w, analyses will be performed with only the post-amendment data (1 mg q4w group: 142 subjects; 1 mg q8w group: 142 subjects; placebo group: 142 subjects). For four null hypotheses, based on multiplicity adjustment based on a gate keeping method using a graphical approach (Figure 8.2.1-1), the power for MT-5547 1 mg SC q4w and 1 mg SC q8w will be 97% and 92% for the primary endpoint, 94% and 87% for the key secondary endpoint, respectively.

Table 3.3-1Change From Baseline at Week 16 in the WOMAC Pain and Physical Function Subscale Scores

| | ] | REGN St | idy R475 | -PN-1227 | | REGN Study R475-PN-0901 | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Placebo<br>(N=83) | MT-5547<br>1 mg<br>(N=85) | MT-5547<br>3 mg<br>(N=84) | MT-5547<br>6mg<br>(N=85) | MT-5547<br>9 mg<br>(N=84) | Placebo<br>(N=55) | MT-5547<br>0.03<br>mg/kg<br>(N=53) | MT-5547<br>0.1<br>mg/kg<br>(N=53) | MT-5547<br>0.3<br>mg/kg<br>(N=54) |
| | Change from baseline in WOMAC pain subscale score | | | | | | | | |
| Baseline | 6.43 | 6.33 | 6.35 | 6.10 | 6.53 | 5.9 | 5.7 | 6.1 | 6.4 |
| n <sup>1)</sup><br>Mean <sup>1)</sup><br>(SD) <sup>1)</sup> | 71<br>-2.43<br>(2.38) | 75<br>-3.49<br>(2.06) | 78<br>-3.39<br>(2.44) | 77<br>-3.07<br>(2.34) | 79<br>-3.81<br>(2.49) | 44<br>-2.4<br>(2.18) | 47<br>-2.7<br>(1.89) | 44<br>-3.4<br>(2.53) | 41<br>-3.2<br>(2.24) |
| LSM <sup>2)</sup> | -2.25 | -3.35 | -3.33 | -3.03 | -3.65 | - | - | - | - |
| Diff. vs. Pbo <sup>3)</sup> | - | -1.10 | -1.08 | -0.78 | -1.40 | - | -0.6 | -1.1 | -0.8 |

| P value | - | 0.0025 | 0.0029 | 0.0304 | 0.0001 | - | 0.1486 | 0.0090 | 0.0488 |
|---|---|---|---|---|---|---|---|---|---|
| | Change f | rom basel | ine in W | OMAC pl | ysical fu | action sub | scale sco | re | |
| Baseline | 6.15 | 6.11 | 6.09 | 5.94 | 6.20 | 5.9 | 5.9 | 6.2 | 6.2 |
| n <sup>1)</sup><br>Mean <sup>1)</sup><br>(SD) <sup>1)</sup> | 70<br>-2.12<br>(2.26) | 75<br>-3.21<br>(2.23) | 78<br>-3.28<br>(2.29) | 76<br>-2.97<br>(2.45) | 80<br>-3.51<br>(2.50) | 44<br>-2.3<br>(2.30) | 47<br>-2.9<br>(1.78) | 44<br>-3.4<br>(2.28) | 41<br>-3.1<br>(2.18) |
| LSM <sup>2)</sup> | -1.98 | -3.08 | -3.27 | -3.03 | -3.41 | - | - | - | |
| Diff. vs. Pbo <sup>3)</sup> | T - | -1.10 | -1.29 | -1.06 | -1.43 | ** | -0.8 | -1.1 | -0.9 |
| P value | - | 0.0019 | 0.0003 | 0.0029 | < 0.0001 | - | 0.0693 | 0.0071 | 0.0245 |

- n: number of subjects at Week 16; mean: arithmetic mean at Week 16; SD: standard deviation at Week 16.
   However, in REGN Study R475-PN-1227, the n includes WOMAC data from after treatment discontinuation.
- 2) LSM: MMRM least squares mean
- 3) Diff. vs. Pbo: Difference for each group relative to the placebo group in the MMRM least squares mean

#### 4. PLANNED ANALYSIS

#### 4.1. Interim Analysis

No interim analysis was planned and hence no multiplicity adjustment for interim analysis is needed.

#### 4.2. Final Analysis

This SAP for 16 week will be finalized before database lock in week 16. The efficacy analysis performed at week 16 is the final efficacy analysis. The analysis for week 16 will be conducted using database up to 16 week after database lock in week 24.

#### 4.3. Independent Data Monitoring Board

An independent data monitoring board will periodically assess unblinded data, and will make recommendations to the study sponsor regarding the appropriateness of continuing the study and about the need for protocol amendments.

The independent data monitoring board will include independent statistical and medical experts. For more details, the overseas independent data monitoring committee procedures (DMC Charter) will be followed.

#### 5. ANALYSIS POPULATIONS

The analysis of efficacy will be performed in the full analysis set (FAS). The principal

analysis set for efficacy will be the modified FAS (mFAS). Secondary analyses of the primary efficacy endpoint and key secondary efficacy endpoint will also be performed in the per-protocol set (PPS). The analysis of safety will be performed in the safety analysis set (SAF). The analysis of pharmacokinetics will be performed in the pharmacokinetic analysis set.

The analysis sets are defined below. For the contents of the data review meeting, refer to a separate materials.

#### (1) Efficacy analysis sets

1) Randomized subjects (RAND)

#### 2) FAS

The FAS will consist of all randomized subjects except for the following subjects.

- Subjects who have not received study drug even once
- Subjects with no WOMAC pain subscale score (the primary endpoint) at baseline
- Subjects with no WOMAC pain subscale score (the primary endpoint) at any time point after randomization

#### 3) Modified FAS (mFAS)

The mFAS will consist of the FAS, except for the following subjects.

- Subjects who are randomized to 3 mg q4w group
- Subjects who are randomized to 6 mg q8w group
- 4) PPS (This set will be used for only statistical analysis for the data obtained from screening to Week 16)

The PPS will consist of the mFAS, except for the following subjects.

- Subjects who did not meet the inclusion criteria
- Subjects who met the exclusion criteria
- Subjects who did not comply with the rules on prohibited concomitant drugs/therapies
- Subjects who did not complete the period from study treatment initiation through the assessment of the WOMAC pain subscale score (the primary endpoint) at Week 16
- Subjects who did not received four injections of study drug

#### (2) SAF

The SAF will consist of all randomized subjects except for the following subjects

- Subjects who did not receive study drug even once
- Subjects for whom absolutely no post-randomization safety data are available

#### 6. STATISTICAL CONSIDERATIONS

#### 6.1. Descriptive Statistics

#### (1) Non-PK related

Continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment group and analysis population being presented, unless otherwise specified.

#### 6.2. Statistical Tests

Unless otherwise specified, all formal statistical tests of treatment effects will be done at two-sided significance level of 0.05. Point estimates will be accompanied with two-sided 95% CIs where applicable.

#### 7. DATA CONVENTIONS

#### 7.1. Analysis Variable Definitions

#### 7.1.1. Study Subjects

#### 7.1.1.1. Demographic and Other Baseline Characteristics

#### (1) BMI

BMI will be recalculated using the formula below and reported to 1dp.

BMI  $(kg/m^2)$  = weight at screening (kg) / {height at screening (m)}<sup>2</sup>

(2) Age(years)

If (month of date of consent > month of date of birth) or (month of date of consent = month of date of birth and day of date of consent >= day of date of birth), then Age (years) = year of date of consent - year of date of birth

if else case, then Age (years) = year of date of consent - year of date of birth -1.

(3) Time since osteoarthritis diagnosis (years)

If (month of date of consent > month of osteoarthritis diagnosis) or (month of date of consent = month of date osteoarthritis diagnosis, and day of date of consent >= day of date of osteoarthritis diagnosis), then Time since osteoarthritis diagnosis (years) = year of date of consent - year of date of osteoarthritis diagnosis

if else case, then Time since osteoarthritis diagnosis (years) = year of date of consent –year of date osteoarthritis diagnosis -1.

Impute date of osteoarthritis diagnosis as the earliest possible date (i.e. first day of month if day is unknown or 1st January if day and month are unknown).

#### 7.1.1.2. Treatment Duration and Compliance

- (1) Treatment Duration
- 1) Treatment Duration (days) = The date of last study drug injection prior to week 16 the date of the first study drug injection + min(28 or (the date of last study drug infection the date of Week 16 study drug injection))
- Criteria for pre-defined limit
   Treatment duration period ≥1 day, ≥29 days, ≥57 days, ≥85 days, and ≥113 days
- (2) Treatment Compliance
- 1) Treatment compliance will be calculated using the formula below and reported to 1dp. Treatment compliance(%) = (Number of injections of study drug during treatment exposure period) / (Number of planned injections of study drug during exposure period on or before the time that the subject discontinues from the study) x = 100%
- 2) Criteria for pre-defined limit the number of injections of study drug: 1, 2, 3 and 4

#### 7.1.2. Efficacy assessments

#### 7.1.2.1. WOMAC pain subscale score

WOMAC pain subscale score

$$= \frac{\text{sum of items from Section A 1 to Section A5 in questionnaire}}{5}$$

#### 7.1.2.2. WOMAC physical function subscale score

WOMAC physical function subscale score

$$= \frac{\text{sum of items from Section C 8 to Section C24 in questionnaire}}{17}$$

#### 7.1.2.3. WOMAC stiffness subscale score

WOMAC stiffness subscale score = 
$$\frac{\text{Section B 6 + Section B7 in questionnaire}}{2}$$

#### 7.1.2.4. WOMAC total score

WOMAC total score

$$= \frac{\text{sum of items from Section A1 to Section C24 in questionnaire}}{24}$$

#### 7.1.2.5. NRS score

- Weekly average walking index joint pain Baseline is defined as the average of the non-missing values during 7 days prior to taking study drug. For each week, the average of the non-missing values during the 7 days on or prior to that week will be used.
- Daily walking index joint pain
   Baseline is defined as the last non-missing values prior to taking study drug.

#### 7.1.2.6. SF-36 / EQ-5D-5L

• SF-36

Physical, Mental and Role social component summary will be calculated considering factor coefficients based on the 1995 Japan National Survey. The derivation of 8 subscales and three component is detailed in appendix 13.1.

EQ-5D-5L
 Utility Index Score will be calculated using the formula and Table below.<sup>[1]</sup>

Utility Index Score

- = 1 + [Estimation of the constant term(if all answer is not 1)]
- + [Sum of "estimation of coefficients corresponding to answer other than 1"]

| Item | Level | Estimation | Standard Error | P-value |
|-----------|-------|------------|----------------|----------|
| Intercept | | - 0.060924 | 0.013625 | < 0.0001 |
| Мо | 2 | -0.063865 | 0.008996 | < 0.0001 |
| | 3 | -0.112618 | 0.009287 | < 0.0001 |
| | 4 | -0.179043 | 0.010231 | < 0.0001 |
| | 5 | -0.242916 | 0.009425 | < 0.0001 |
| Sc | 2 | -0.043632 | 0.008931 | < 0.0001 |
| | 3 | - 0.076660 | 0.009972 | < 0.0001 |
| | 4 | - 0.124265 | 0.010129 | < 0.0001 |
| | 5 | - 0.159659 | 0.008924 | < 0.0001 |
| | 2 | -0.050407 | 0.009205 | < 0.0001 |
| | 3 | -0.091131 | 0.010005 | < 0.0001 |
| Ua | 4 | -0.147929 | 0.009744 | < 0.0001 |
| | 5 | -0.174786 | 0.009115 | < 0.0001 |
| Pđ | 2 | - 0.044545 | 0.008354 | < 0.0001 |
| | 3 | -0.068178 | 0.010052 | < 0.0001 |
| | 4 | -0.131436 | 0.008985 | < 0.0001 |
| | 5 | -0.191203 | 0.009604 | < 0.0001 |
| Ad | 2 | -0.071779 | 0.009701 | < 0.0001 |
| | 3 | -0.110496 | 0.010863 | < 0.0001 |
| | 4 | -0.168171 | 0.009850 | < 0.0001 |
| | 5 | -0.195961 | 0.009164 | < 0.0001 |

Mo: mobility, Sc: self-care, Ua: usual activities, Pd: pain/discomfort, Ad: anxiety/depression

e.g ) If answer is [1 1 1 1 1], Utility Index Score is = 1+0+0=1. If answer is [1 1 3 2 1], Utility Index Score is = 1+(-0.060924)+(-0.091131-0.068178)=0.779767.

#### 7.1.2.7. Response rate based on the OMERACT-OARSI criteria



Note that the criteria in the diagram above are based on standardized score between 0 and 100. For this study, WOMAC pain and physical function subscale score are between 0 and 10, so the absolute change required for response is the required change in the diagram above divided by 10; PGA is 1, 2, 3, 4 or 5, so the absolute change required for response is at least 1 point.

#### 7.1.2.8. Rescue Medication

Baseline amount of rescue medication use is defined as the average of the non-missing values during 7 days prior to taking study drug. For each week, the average of the non-missing values during the 7 days on or prior to that week will be used.

#### 7.1.3. Safety Assessments

The on-treatment period is defined as the time from first dose of investigational product up to 28 days after the last dose of investigational product excluding adverse events after study drug sc administration at week 16.

#### 7.1.3.1. Adverse Events

Adverse events will be coded according to the MedDRA version 20.1

(1) Treatment Emergent Adverse Events/ Treatment Emergent Serious Adverse Events (TEAEs/TESAEs)

An AE/SAE is classified as treatment emergent if it newly occurred after the first dose of study drug or if a pre-dose event increases in severity following the first dose of study drug.

(2) Adverse Drug Reaction

A TEAE is considered "adverse drug reaction" if it has been assessed as having a "reasonable

possibility" in relationship to the study drug.

#### (3) Adverse Event of Special Interest(AESI)

Adjudicated arthropathy, sympathetic nerve disorders and altered peripheral sensation are defined as adverse events of special interest (AESI) to facilitate characterizing the safety profile of MT-5547.

#### (4) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1

#### 7.2. Analysis Visit Definitions

#### (1) General analysis visit definitions

| Analysis visit | Nominal day | Window |
|----------------|-------------|-------------------------|
| Baseline | Day 1 | <day 1<="" td=""></day> |
| Week 1 | Day 8 | Day 2 to 11 |
| Week 2 | Day 15 | Day 12 to 21 |
| Week 4 | Day 29 | Day 22 to 43 |
| Week 8 | Day 57 | Day 44 to 71 |
| Week 12 | Day 85 | Day 72 to 99 |
| Week 16 | Day 113 | Day 100 to 127 |

#### (2) For NRS analisys visit definitions

| Analysis visit | Window |
|----------------|----------------|
| Baseline | Day -7 to -1 |
| Week 1 | Day 1 to 7 |
| Week 2 | Day 8 to 14 |
| Week 3 | Day 15 to 21 |
| Week 4 | Day 22 to 28 |
| Week 5 | Day 29 to 35 |
| Week 6 | Day 36 to 42 |
| Week 7 | Day 43 to 49 |
| Week 8 | Day 50 to 56 |
| Week 9 | Day 57 to 63 |
| Week 10 | Day 64 to 70 |
| Week 11 | Day 71 to 77 |
| Week 12 | Day 78 to 84 |
| Week 13 | Day 85 to 91 |
| Week 14 | Day 92 to 98 |
| Week 15 | Day 99 to 105 |
| Week 16 | Day 106 to 112 |

The date of the first dose of study drug is defined as Day 1.

Unless otherwise specified, baseline will be the last observed value of the parameter of

interest prior to the first intake of study drug (this includes unscheduled visits). For other visits, if there are multiple data in a window, the closest data to nominal day will be used. If the distance to the nominal day is the same, the data of later date will be used.

#### 7.3. Data Handling Convention for Missing Data

#### (1) Non-PK related

Efficacy:

#### **WOMAC**

WOMAC scores will be computed when one pain, one stiffness, or 1-3 physical function items are missing. The missing items will be imputed by the mean of available items within the same subscale. The scores will be set to missing if more items are missing.

#### **NRS**

If all values are missing for the 7 days, the value for that week is set to missing.

#### SF-36 / EQ-5D-5L

- SF-36 subscale scores will be computed if at least 50% of items are available. The missing items will be imputed by the mean of available items.
- EQ-5D-5L index will be set to missing if any of the 5 dimensions is missing.

#### Adverse events:

If severity or relationship is found to be missing the most severe occurrence will be imputed for the summary of interest.

For AE start missing or partial dates, the AE will be treated as TEAE if it cannot be determined to be a non-TEAE.

#### 8. STATISTICAL METHODOLOGY

#### 8.1. Study Subjects

#### 8.1.1. Subject Disposition

Subject disposition will be summarized by treatment group, combined MT-5547 and overall on the randomized population.

#### 8.1.2. Analysis Populations

Analysis populations will be summarized by treatment group, combined MT-5547 and overall on the randomized population.

#### 8.1.3. Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | category | Descriptive |
|---|---|---|
| Sex | Male, Female | |
| Age(years) | <65,>=65 | Yes |
| Height(cm) | | Yes |
| Weight(kg) | - | Yes |
| BMI(kg/m2) | <25, >= 25 and < 30,<br>>=30 | Yes |
| Race | Japanese, other | |
| Time since OA diagnosis (years) | <1, >=1 and <5, >=5<br>and <10, >=10 | Yes |
| Index Joint | Knee, Hip | |
| K-L score for index joint | 1, 2, 3, 4 | |
| WOMAC pain subscale score | <6,>=6 | Yes |
| WOMAC Physical function subscale score | <6,>=6 | Yes |
| PGA | 1, 2, 3, 4, 5 | Yes |
| Pain site | Right Knee, Left<br>Knee, Right Hip, Left<br>Hip, Right Shoulder,<br>Left Shoulder | |
| Pretreatment drug | NSAIDs(Systemic use), NSAIDs(Topical use), Acetaminophen, Opioid, Monoamine reuptake inhibitor, Hyaluronic acid, Pregabalin, Herbal medicine, Other | |
| NSAIDs Inadequate Pain Relief | Yes, No | |
| NSAIDs Intolerance | Yes, No | |
| Ever taken Opioid for Pain due to OA | Yes, No | |
| Opioid Inadequate Pain<br>Relief | Yes, No | |
| Opioid Intolerance | Yes, No | |
| Ever taken Acetaminophen for Pain due to OA | Yes, No | |
| Acetaminophen | Yes, No | |

| Inadequate Pain Relief | |
|-------------------------------------------------------------|---------|
| Acetaminophen<br>Intolerance | Yes, No |
| NSAID + Opioid +<br>Acetaminophen<br>Inadequate Pain Relief | Yes, No |

Demographic and other baseline characteristics will be summarized by treatment group, combined MT-5547 and overall on the FAS population, PPS population and the SAF population.

Demographic and other baseline characteristics before the protocol amendment and after the protocol amendment will be summarized by treatment group, combined MT-5547 and overall on the mFAS population.

#### 8.1.4. Treatment Duration and Compliance

Treatment duration will be summarized by treatment group and combined MT-5547 on the SAF population. Treatment compliance will be summarized by treatment group and combined MT-5547 on the SAF population.

#### 8.2. Efficacy Assessments

Efficacy assessment will be summarized by treatment group on the mFAS population.

#### 8.2.1. Primary Efficacy Endpoint

The change in the WOMAC pain subscale score from baseline to Week 16 will be summarized and plotted by treatment group.

#### Primary analysis method

The primary analysis will be tested using the estimator of mixed effect model for repeated measurement (MMRM) approach. The model will include the treatment group, measurement time point, treatment group and measurement time point interaction, stratification factor K-L grade (2-3 or 4), and stratification factor evaluated joint (knee or hip) as factors, and the baseline and baseline and measurement time point interaction as covariates. The within-subject correlation structure will be unstructured, and the denominator degrees of freedom for the test statistics of estimated parameters will be approximated using the Kenward-Roger method. In case the model will not converge with the unstructured covariance structure, Heterogeneous Autoregressive (1) (ARH[1]), Heterogeneous Compound Symmetry (CSH), Autoregressive (1) (AR[1]) or Compound Symmetry(CS) covariance structure will be used instead in this order.

#### • Evaluation on 1 mg q4w group

With pooling the data on 1 mg q4w and placebo obtained before and after the protocol amendment (Ver. 04.00.00000), the least square mean, standard error, P value, and 95% confidence interval of the difference between each of the MT-5547 1 mg q4w and the placebo group in the change in the WOMAC pain subscale score from baseline to Week 16 will be calculated using the MMRM approach.

#### • Evaluation on 1 mg q8w group

Using only the data obtained after the protocol amendment (Ver. 04.00.0000), the least square mean, standard error, P value, and 95% confidence interval of the difference between each of the MT-5547 1 mg q4w, MT-5547 1 mg q8w and the placebo groups in the change in the WOMAC pain subscale score from baseline to Week 16 will be calculated using the MMRM approach.

MMRM that assumes that the missing mechanism is missing at random (MAR) is an analysis method in which missing values are not replaced. This model will be used to estimate the treatment effect in the mFAS when subjects continue receiving treatment through Week 16.





#### Sensitivity analyses

Sensitivity analysis will use the same estimator as for the primary analysis. Likelihood based model method on the mFAS under Missing Not at Random(MNAR) assumption will be performed using the same MMRM as specified for the primary analysis. The following additional analyses will be performed for the primary efficacy endpoint.
#### • Multiple Imputation (MI) analysis by Reason for Discontinued Treatment

The missing data for patients who discontinued treatment due to lack of efficacy or AEs will be imputed with values centered at the mean baseline value of the treatment group that patients were randomized to. The missing data for patients discontinued treatment due to other reasons will be imputed under missing-at-random assumption using the regression method with adjustment for covariates including treatment group, randomization strata, and baseline score. Intermittently missing data will be imputed using Markov Chain Monte Carlo method.

The primary efficacy variables will be analyzed using a multiple imputation approach with mixed-effect model for repeated measure (MMRM) based on the mFAS with adjustment for missing data due to treatment discontinuation for the reasons of lack of efficacy or AEs assuming the WOMAC scores would on average return to baseline values. Missing data up to week 16 will be imputed 50 times to generate 50 complete data sets by using the SAS procedure PROC MI following the 4 steps below:

Step 1: This methodology will structure data based on missing data patterns. The Pattern Mixture Model (PMM) method will be based on a missingness pattern having a monotone structure, i.e. if among the observations over time one data value is missing, all other values after this missing value will also be missing. For patients with intermittent missing values, before performing MI based on the PMM, it will be necessary to create a monotone missingness pattern. Intermittent missing values will be imputed using the Markov Chain Monte Carlo (MCMC) methodology which assumes a multivariate normal distribution over all variables included in the imputation model. The MI procedure in SAS will be used for this purpose and this first MI step is planned to be repeated 50 times, creating different datasets with a monotone missing data structure. Seed value of 1995 will be used in the MI procedure. The imputation is based on the MAR assumption, i.e. the missing data are assumed to follow the same model as the other patients in their respective treatment group.

The following SAS code will be used to generate the monotone missing data pattern:



Step 2: After this, the remaining missing data will be imputed using a method for monotone missingness, also based on the MAR assumption. Thus, for each of the created dataset with a monotone missing data pattern, the MI procedure in SAS will be used to impute missing values within the instrument range based on a sequential procedure reflecting the monotone missing data pattern. Patients with the first missing value occurring at Week 1 ('W1') will have their missing Week 1 value replaced by an imputed value from a regression model with treatment group ('TRTP'), K-L grade ('GRADE'), index joint ('INDEX') and baseline ('BASE') value as explanatory variables. In the next step, patients with their Week 2 ('W2') value missing will have their missing Week 2 value replaced by an imputed value from a regression model with treatment group, grade, index and baseline and the Week 1 value as explanatory variables. Similar procedure will be used to replace the missing values at Week 4, Week 8, Week 12 and Week 16.

The following SAS code will be used to make the imputation with the MAR assumption:



<u>Step 3</u>: The initially missing and now imputed data for patients discontinued from the study treatment due to lack of efficacy or AEs will be adjusted to be centered at the mean baseline value for that treatment group, i.e., final imputed score = imputed score under MAR - (mean change from baseline score at the post-baseline time point\* for the treatment group based on patients on treatment with non-missing data at that time point).

\* MMRM models similar to that described for the primary analysis will be run on each of the 50 generated imputed datasets and the differences between the treatment groups at the

post-baseline time point.

Step 4: The imputed datasets generated with the approach described above do contain only non-missing values and are used as input in the model for the sensitive analysis for the primary efficacy endpoint. Any score imputed outside the range of the WOMAC subscale score of 0-10 will be truncated to the nearest permissible value on the WOMAC scale. MMRM models similar to that described for the primary analysis will thus be run on each of the 50 generated imputed datasets and the differences between the treatment groups at Week 16 of the DBDD Maintenance period will be estimated (and export to data 'ESTIMATES'). Finally, the MIANALYZE procedure in SAS will be applied to combine the results from these analyses to derive an overall estimate of the treatment differences at W16 according to the following code. In addition to the estimates, corresponding 95% confidence intervals and p-values will be calculated.

#### • Tipping Point Analysis with MNAR assumption

Sensitivity analysis using a tipping point approach with multiple imputation will be performed to assess the robustness of the results due to data that may be missing not-at-random (MNAR).

This approach will introduce a sensitivity parameter,  $\delta$ . Estimations will be performed using multiple imputation methodology. Missing data up to week 16 time point will be imputed 50 times to generate 50 complete datasets by using SAS procedure PROC MI for each  $\delta$  following the 3 steps below:

Step 1 and 2: The same as step 1 and 2 for Multiple Imputation (MI) analysis by Reason for Discontinued Treatment. The imputation is based on the MNAR assumption, not based on the MAR assumption. Any score imputed outside the range of the WOMAC subscale score of 0-10 will be truncated to the nearest permissible value on the WOMAC scale.

The following SAS code will be used to make the imputation with the MNAR assumption:



Step 3: Each imputed data set will be analyzed using the MMRM model with treatment, randomization strata, and relevant baseline included in the model. For each  $\delta$  the SAS MIANALYZE procedure will be used to generate valid statistical inferences by combining results from the 50 analyses using Rubin's formula. By progressively increasing  $\delta$ , the sensitivity analysis will explore the tipping points, e.g.,  $\delta$  value when the p-value for a treatment comparison is above 0.05. Results will be then summarized using summary tables and graphs.

#### Multiplicity adjustment

Because this study is a confirmatory study, in order to keep the family wise type 1 error rate to a significance level of 5% (alpha), two-sided, in the tests of the following hypotheses regarding the primary endpoint and the key secondary efficacy endpoint, a gatekeeping method based on a graphical approach will be used to perform multiplicity adjustment, as shown in Figure 8.2.1-1 to verify the hypotheses (Bretz et al., 2009). This multiplicity adjustment will only be performed for the statistical analyses of data from the double-blind period from screening to Week 16 after treatment initiation.

- Null hypothesis H01: The change from baseline in the WOMAC pain subscale score at Week 16 in the 1 mg SC q4w group is the same as that in the placebo group
- Null hypothesis H02: The change from baseline in the WOMAC pain subscale score at

Week 16 in the 1 mg SC q8w group is the same as that in the placebo group

- Null hypothesis H03: The change from baseline in the WOMAC physical function subscale score at Week 16 in the 1 mg SC q4w group is the same as that in the placebo group
- Null hypothesis H04: The change from baseline in the WOMAC physical function subscale score at Week 16 in the 1 mg SC q8w group is the same as that in the placebo group



Figure 8.2.1-1: MT-5547 Multiple Test Procedure

#### Subgroup analysis

Subgroup analyses will be performed on the primary endpoint. Each subgroup is following at baseline timepoint:

- index joint (hip or knee)
- K-L score category(2-3 or 4)
- WOMAC pain (<6 or >=6)
- OA Duration(<5 or >=5)
- age (<65 or >=65)
- sex(Male, Female)
- BMI (<25 or >=25)
- Weight(<median or >=median)
- Opioid (Yes or No)

Each subgroup will be analyzed separately for the primary endpoint using MMRM model similar to the primary model.

Change from baseline to week 16 for the subgroup of index joint (hip or knee) and K-L score category(2-3 or 4) will be summarized by visit. Change from baseline to week 16 for the other subgroup will be summarized at week 16. In addition, forest plot depicting the treatment effect, p-values for interaction terms between the treatment group and each subgroup and 95% CI for each subgroup will be displayed.

#### Supplemental analysis

The PPS will be analyzed using the same method as for the primary analysis to confirm the robustness of the results of the primary analysis for the effects of the analysis set.

#### Supplementary analysis with respect to the data pooling on 1 mg q4w and placebo

The data on 1 mg q4w and placebo obtained before and after the protocol amendment (Ver. 04.00.00000) will be analyzed using the same method as for the primary analysis to confirm the data homogeneity and the robustness of the results of the primary analysis. Also, homogeneity in demographic and other baseline characteristics [Section 8.1.3] between data obtained before and after the protocol amendment will be confirmed.

#### Supplementary analysis with respect to response the site differences

Absolute values and changes from baseline will be summarized at week 16 by treatment group and site.

#### 8.2.2. Key Secondary Efficacy Endpoints

The change in the WOMAC physical function subscale score from baseline to Week 16 will be analyzed on the mFAS and PPS population as the key secondary endpoint using the same primary analysis method (MMRM) and same subgroup analysis and supplementary analysis with respect the data pooling on 1mg q4w and placebo will be performed. Multiplicity adjustment described in Section 8.2.1.

#### 8.2.3. Other Efficacy Endpoints

### WOMAC pain subscale score, WOMAC physical function subscale score, WOMAC stiffness subscale score, WOMAC total score, WOMAC individual score and PGA

For the changes from baseline at each visit in the WOMAC pain subscale score, the WOMAC physical function subscale score, the WOMAC stiffness subscale score, the WOMAC total score, WOMAC individual score and PGA, the same primary analysis method (MMRM) described in Section 8.2.1 will be analyzed. And the WOMAC pain subscale score will also be summarized at each visit by treatment group on the FAS population. In addition,

change from baseline to week 16 in WOMAC pain subscale score, WOMAC physical function subscale score and PGA will be graphed by visit.

#### Weekly average and daily walking index joint pain using NRS

For the change from baseline in the weekly average and daily walking index joint pain using NRS, the same primary analysis method (MMRM) described in Section 8.2.1 will be analyzed. In addition, change from baseline to week 16 in weekly average walking index joint pain using NRS will be graphed by visit.

#### SF-36 / EQ-5D-5L

For the changes from baseline at each visit in SF-36 eight subscale summary scores and three component summary socres / EQ-5D-5L visual analogue scale(VAS) and utility index scores, the same primary analysis method (MMRM) described in Section 8.2.1will be analyzed.

## <u>Proportions of subjects with improvement of 30%, 50%, 70% and 90% at each visit compared to baseline in WOMAC pain subscale score, WOMAC physical function subscale score and PGA</u>

A generalized linear mixed-effects model (GLMM) by logit type for response variable will be used to evaluate these binary response variables. The denominator degrees of freedom for the test statistics of estimated parameters will be approximated using the Kenward-Roger method. The estimated response rate for each treatment group and placebo group, P value, and 95% confidence interval of the odds ratio of each of the MT-5547 1 mg q4w and MT-5547 1 mg q8w groups compared to the placebo group in each binary response variables will be calculated at each visit using this GLMM approach.

- The covariates: baseline and the interaction of baseline and measurement time point.
- The fixed factors: Treatment group, measurement time point, the interaction of treatment group and measurement time point, K-L grade (2-3 or 4), and evaluated joint location (knee or hip)
- Random factors: Intercept for subject

The SAS code planned for the analysis is outlined below.



## Response rate based on the OMERACT-OARSI criteria at Week 16 compared to baseline

Responder analyses for OMERACT-OARSI will be summarized at each visit using the same GLMM approach in previous model.

#### Proportion subjects who used rescue medication

The proportion of subjects taking rescue medication in baseline and up to week 16 will be summarized by treatment group. Number of days on rescue medication during treatment priod(Day1 to Day 28, Day 29 to Day 56, Day 57 to Day 84, Day 85 to Day 112) will be summarized by treatment group. Number of weekly average usage of rescue medication will be summarized at each week by treatment group.

#### 8.3. Safety Assessments

Safety assessments will be made on the SAF population.

#### 8.3.1. Adverse Events

Overall summary for the following will be conducted.

- Subjects with at least one TEAE
- Subjects with at least one adverse drug reaction
- Subjects with at least one TESAE
- Subjects with at least one serious adverse drug reaction
- Subjects with at least one AESI
- Subjects with at least one TEAE leading to discontinuation of study drug
- Subjects with TEAE leading to death

The following summaries also will be conducted.

- TEAEs by SOC and PT
- Adverse drug reactions by SOC and PT
- AESI by SOC and PT
- TESAEs by SOC and PT
- Serious adverse drug reactions by SOC and PT
- TEAEs leading to discontinuation of study drug by SOC and PT
- TEAEs by SOC, PT and severity
- Adverse drug reactions by SOC, PT and severity

Each of the summaries will be done by treatment group at the subject level - multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the

maximum severity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility/no reasonable possibility) and/or the earliest duration.

#### 9. DATA PRESENTATION CONVENTIONS

#### 9.1. Number of Digits to Report

#### (1) Non-PK related

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as the data provided in the datasets | All original (i.e. non-derived) |
| | see section 7.3 | All derived data |
| Mean, Median, SD, SE,<br>Confidence intervals | One more DP than above | All |
| Percentages*1 | 1 DP | All |
| Ratios | 3 DPs | All |
| p-values*2 | 3 DPs | All |

<sup>\*1</sup> Percentages: use 1 place beyond the decimal point, except for the following cases:

If the percentage is equal to 0, then leave blank, do not use (0)

If the percentage is equal to 100, then use "(100)" without a decimal

If the p-value is less than 0.001, then use p<0.001

#### 9.2. Treatments to Report

| For TFLs |
|------------------|
| MT-5547 1 mg q8w |
| MT-5547 1 mg q4w |
| MT-5547 Combined |
| MT-5547 3 mg q4w |
| MT-5547 6 mg q8w |
| Placebo |
| Total |

#### 9.3. Analysis Visits to Report

#### (1) Non-PK related

Efficacy:

| Analysis Visit | Apply to | | | |
|---|---|---|---|---|
| | WOMAC and PGA | SF-36 and<br>EQ-5D-5L | Weekly<br>average NRS<br>and Rescue | Daily NRS |

<sup>\*2</sup> p-values: use 3 places beyond the decimal point, except for the following cases:

| | | | Medicine | |
|----------|---|---|----------|---|
| Baseline | X | X | X | X |
| Day 1 | | | | X |
| Day 2 | | | | X |
| Day 4 | | | | X |
| Day 6 | | | | X |
| Week 1 | X | | X | X |
| Week 2 | X | | X | X |
| Week 3 | | | X | X |
| Week 4 | X | X | X | X |
| Week 5 | | | X | X |
| Week 6 | | | X | X |
| Week 7 | | | X | X |
| Week 8 | X | X | X | X |
| Week 9 | | | X | X |
| Week 10 | | | X | X |
| Week 11 | | | X | X |
| Week 12 | X | | X | X |
| Week 13 | | | X | X |
| Week 14 | | | X | X |
| Week 15 | | | X | X |
| Week 16 | X | X | X | X |

#### 10. CHANGE FROM THE PROTOCOL

There are currently no changes to analysis from protocol.

#### 11. SOFTWARE

All statistical analyses will be performed using SAS version 9.3 or higher.

#### 12. REFERENCES

- [1] Shinya I, Takeru S, Ataru I, Shinichi N, Takashi F, et al. Developing a Japanese version of the EQ-5D-5L value set. J. Natl. Inst. Public Health.2015;64 (1): 47-55.
- [2] Fukuhara S, Suzukamo Y. Manual of SF-36v2 Japanese version: Institute for Health Outcomes & Process Evaluation research. Kyoto: 2004. Ver3/2011.

#### 13. APPENDIX

#### 13.1. SF-36v2 Scoring Algorithm<sup>[2]</sup>











# Statistical Analysis Plan (For Database at Week 68)


A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study on MT-5547 in Patients with Osteoarthritis Accompanied by Moderate to Severe Pain

| Prepared By: | Mitsubishi Tanabe Pharma Corporation |
|--------------|--------------------------------------|
| Version: | 1.0 |
| Date: | 19-April-2021 |

#### APPROVAL FORM

#### Statistical Analysis Plan(For Database at Week 68)

|---|---|
| Protocol Title | A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study<br>on MT-5547 in Patients with Osteoarthritis Accompanied by<br>Moderate to Severe Pain |
| Version / Date | 1.0 / 19-April-2021 |

#### Authors:

| Statistics Author | |
|-------------------|-------------------|
| Print Name: | |
| Position: | Biostatistician |
| Clinical Pharmac | cokinetics Author |
| Print Name: | |
| Position: | Pharmacokinetics |

#### Approved by:

| Statistic Approver | |
|--------------------|------------------------------|
| Print Name: | |
| Position: | Responsible Biostatistician |
| Signature: | Refer to email |
| Approval date: | Refer to email |
| Clinical Pharmaco | kinetic Approver |
| Print Name: | |
| Position: | Responsible Pharmacokinetics |
| Signature: | Refer to email |
| Approval date: | Refer to email |

#### TABLE OF CONTENTS

| 1. | INTRODUCTION | 8 |
|---|---|---|
| 2. | STUDY OBJECTIVE AND ENDPOINTS | 8 |
| | 2.1. Study Objective(s) | 8<br>9 |
| 3. | STUDY DESIGN | 10 |
| | <ul> <li>3.1. Study Design</li> <li>3.2. Schedule of Study Procedures</li> <li>3.2.1. Test/Observation Schedule</li> <li>3.3. Sample Size and Power Considerations</li> </ul> | 11<br>11 |
| 4. | PLANNED ANALYSIS | 19 |
| | <ul> <li>4.1. Interim Analysis</li> <li>4.2. Final Analysis</li> <li>4.3. Independent Data Monitoring Board</li> </ul> | 19 |
| 5. | ANALYSIS POPULATIONS | 19 |
| 6. | STATISTICAL CONSIDERATIONS | 21 |
| | 6.1. Descriptive Statistics | |
| 7. | DATA CONVENTIONS | 21 |
| | 7.1. Analysis Variable Definitions 7.1.1. Study Subjects 7.1.1.1. Demographic and Other Baseline Characteristics 7.1.1.2. Medical History 7.1.1.3. Prior or Concomitant Medication 7.1.1.4. Treatment Duration, Treatment and Post-Treatment Ob | 21<br>22<br>23<br>oservation |
| | Duration and Compliance | |
| | <ul> <li>7.1.2.1. WOMAC pain subscale score</li></ul> | 24<br>24<br>24 |
| | 7.1.2.5. SF-36 / EQ-5D-5L | 24 |
| | <ul><li>7.1.2.6. Response rate based on the OMERACT-OARSI criteria</li><li>7.1.2.7. Rescue Medication</li></ul> | 26<br>26 |

| | 7.1.3. Safety Assessments | 26 |
|---|---|---|
| | 7.1.3.1. Adverse Events | |
| | 7.1.3.2. Laboratory Tests | 28 |
| | 7.1.3.3. Vital Signs | |
| | 7.1.3.4. ECG 29 | |
| | 7.1.4. Pharmacokinetics Evaluation | 29 |
| | 7.1.4.1. MT-5547 Concentrations in Serum | 29 |
| | 7.1.4.2. Anti-Drug Antibodies in Serum | 29 |
| | Analysis Visit Definitions | 30 |
| | 7.2. 30 | |
| | 7.3. Data Handling Convention for Missing Data | 32 |
| 8. | STATISTICAL METHODOLOGY | 33 |
| | 8.1. Study Subjects | 33 |
| | 8.1.1. Subject Disposition | |
| | 8.1.2. Analysis Populations | 33 |
| | 8.1.3. Site Enrollment | 33 |
| | 8.1.4. Demographic and Other Baseline Characteristics | 33 |
| | 8.1.5. Medical History | 35 |
| | 8.1.6. Radiograph eligibility data | 35 |
| | 8.1.7. Prior or Concomitant Medications | 35 |
| | 8.1.8. Treatment Duration, Treatment and Post-Treatment Observation Duration | on and |
| | Compliance | 35 |
| | 8.2. Efficacy Assessments | |
| | 8.2.1. Other Efficacy Endpoints | 35 |
| | 8.2.2. Assessment of self-injection | |
| | 8.3. Safety Assessments | |
| | 8.3.1. Adverse Events | |
| | 8.3.2. Laboratory Tests | 40 |
| | 8.3.3. Vital Signs | |
| | 8.3.3.1. Assessment of Orthostatic Blood Pressure with standing value | |
| | supine value | 41 |
| | 8.3.4. ECGs 41 | 42 |
| | 8.3.5. Physical Examinations | |
| | · | |
| | 8.3.7. JOA score | |
| | 8.3.9. Injection Site Assessments | 42<br>43 |
| | 8.3.10. Autonomic Symptoms Questionnaire | 43 |
| | 8.3.11. Neurological Examinations | 43 |
| | 8.3.12. Joint Pain Questionnaire | |
| | 8.3.13. Joint Replacement | 44 |
| | 8.4. Pharmacokinetics Evaluation | 44 |
| | 8.4.1. Analysis of Anti-Drug Antibody in Serum | |
| | 8.4.2. Assessment of Concentration-Response Relationships | 45 |
| | 8.4.3. | 45 |
| 9. | DATA PRESENTATION CONVENTIONS | |

| Statistical Analysis Plan<br>Protocol No. MT-5547-J01 | | | Mitsubishi Tanabe Pharma Corporation |
|---|---|---|---|
| | | | 45<br>46 |
| | 9.2.<br>9.3. | 46 Analysis Visits to Report | 46 |
| 10. | CHAI | NGE FROM THE PROTOCOL | 49 |
| 11. | . SOFTWARE | | 49 |
| 12. | 2. REFERENCES | | 49 |

#### **ABBREVIATIONS**

| Abbreviations | Definitions |
|---------------|-------------------------------------------------------------|
| ADA | anti-drug antibodies |
| AE | adverse event |
| AESI | Adverse event of special interest |
| ALP | alkaline phosphatase |
| ALT | alanine transaminase |
| ANCOVA | analysis of covariance |
| AST | aspartate transaminase |
| ATC | anatomical therapeutic chemical |
| BAP | bone specific alkaline phosphatase |
| BDR | blinded data review |
| BLQ | below limit of quantification |
| BMI | body mass index |
| CI | confidence interval |
| CRP | C-reactive protein |
| CV | coefficient of variation |
| DA | destructive arthropathy |
| DBP | diastolic blood pressure |
| DMC | data monitoring committee |
| DP | decimal places |
| ECG | 12-lead electrocardiogram |
| EQ-5D-5L | EuroQol-5-Domain-5-Level health questionnaire |
| FAS | full analysis set |
| K-L | Kellgren-Lawrence |
| LLOQ | lower limit of quantification |
| MAR | missing at random |
| MedDRA | medical dictionary for regulatory activities |
| MMRM | mixed effect model for repeated measures |
| NAb | neutralizing anti-drug antibody |
| NGF | nerve growth factor |
| NRS | numerical rating scale |
| NSAID | nonsteroidal anti-inflammatory drug |
| OA | osteoarthritis |
| OMERACT- | Outcome Measures in Rheumatology Arthritis Clinical Trials- |
| OARSI | Osteoarthritis Reseach Society International |
| PD | pharmacodynamics |
| PGA | patient global assessment |
| PK | pharmacokinetics |
| PR | pulse rate |
| PT | MedDRA preferred term |
| Q4W | every 4 weeks |
| Q8W | every 8 weeks |

| QOL | quality of life |
|-------|---------------------------------------------------|
| RAND | all subjects randomized population |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SC | subcutaneous |
| SD | standard deviation |
| SF-36 | Short Form 36-item health survey |
| SIF | Subchondral insufficiency fracture |
| SOC | system organ class |
| TEAE | treatment emergent adverse event |
| TESAE | treatment emergent serious adverse events |
| ULN | upper limit of normal range |
| WHO | World Health Organization |
| WOMAC | Western Ontario and McMaster Osteoarthritis Index |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol (v4.0) dated 31-July-2018. This protocol will plan to respectively perform the statistical analysis for the clinical trial data from screening to Week 16, from screening to Week 24 and from screening to Week 68.

For the clinical trial data from screening to Week 68, this SAP covers statistical analysis, tabulations and listings of the study data to investigate the efficacy and safety of MT-5547 SC 1mg q4w and 1mg q8w compared to matching placebo. Therefore, this SAP will be finalized prior to database lock at Week 68 to ensure the credibility of the study results by pre-specifying the statistical methods for the data analyses before un-blinding of treatment assignments. For the clinical trial data from screening to Week 16 and from screening to Week 24 was separately created.

Any statistical analysis details described in this document supersede any description of statistical analysis in the protocol.

#### 2. STUDY OBJECTIVE AND ENDPOINTS

#### 2.1. Study Objective(s)

The objective of this study is to verify the superiority of 16 weeks of MT-5547 treatment to placebo, as evidenced by the WOMAC pain subscale score (the efficacy outcome measure), in patients with osteoarthritis of the knee or hip. Additional objectives of the study are to investigate the efficacy, safety, and pharmacokinetics of MT-5547 in long-term use.

#### 2.2. Study Endopoint(s)

#### 2.2.1. Efficacy Endpoint(s)

- (1) Primary efficacy endpoint
  WOMAC pain subscale score (change from baseline at Week 16)
- (2) Key secondary efficacy endpoint
  WOMAC physical function subscale score (change from baseline at Week 16)
- (3) Secondary efficacy endpoints
  - 1) Patient global assessment (PGA) (change from baseline at each assessment time point)
  - 2) WOMAC pain subscale score (change from baseline at each assessment time point)
  - 3) WOMAC physical function subscale score (change from baseline at each assessment time point)
  - 4) WOMAC stiffness subscale score (change from baseline at each assessment time point)
  - 5) WOMAC total score (change from baseline at each assessment time point)
  - 6) Proportions of subjects with 30%, 50%, 70% and 90% improvements in their WOMAC pain subscale scores compared to baseline (at each assessment time point)

- 7) Proportions of subjects with 30%, 50%, 70% and 90% improvements in their WOMAC physical function subscale scores compared to baseline (at each assessment time point)
- 8) Proportions of subjects with 30%, 50% and 70% improvements in their PGA compared to baseline (at each assessment time point)
- 9) Numerical Rating Scale (NRS) score for the mean pain on walking in the evaluated joint (change from baseline at each assessment time point)
- 10) SF-36 (change from baseline at each assessment time point)
- 11) EQ-5D-5L (change from baseline at each assessment time point)
- 12) Improvement rate based on the Outcome Measures in Rheumatology Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) criteria (at each assessment time point)
- 13) Amount of rescue medication used (number of days on which rescue medication was used, and amount [number of tablets] used)

#### 2.2.2. Safety Assessment(s)

- (1) Adverse events and adverse reactions (clinically significant adverse events were identified as being adjudicated arthropathy, sympathetic nervous system disorders and altered peripheral sensation)
- (2) General clinical laboratory tests
- (3) Body weight
- (4) Vital signs
- (5) ECG
- (6) Physical examination
- (7) Joint pain questionnaire
- (8) Survey of autonomic symptoms
- (9) Assessment of orthostatic blood pressure
- (10) Neurological assessments
- (11) Bone density
- (12) Imaging Tests
- (13) Injection site assessments
- (14) Assessments of subjects undergoing joint replacement

#### 2.2.3. Pharmacokinetics Assessment(s)

MT-5547 concentration in serum

Anti-MT-5547 antibody in serum

#### 2.2.4. Pharmacodynamics Endpoint(s)

Efficacy: WOMAC pain subscale score, WOMAC physical function subscale score, PGA Safety: alkaline phosphatase (ALP), C-reactive protein (CRP), bone specific alkaline phosphatase (BAP)

#### 3. STUDY DESIGN

#### 3.1. Study Design

Study Phase: Phase 2/3

Type of Study: Confirmatory Study

Parallel group, randomized, placebo-controlled, double-blind (24 weeks), multicenter





- 1) The post-treatment observation period will be the 20 weeks from the day after the end of the 48-week treatment period. Furthermore, for subjects discontinued from the study, the post-treatment observation period will be the 24 weeks from the administration of MT-5547 or MT-5547 placebo. If a joint replacement procedure is going to be performed, the postoperative test observation period will be the period from the day after the day of discontinuation until 20 weeks after the joint replacement procedure is performed.
- 2) From Week 16 to Week 48, the placebo group will receive an additional dose of naproxen tablets to reduce the dropout rate in the placebo group. The MT-5547 group will receive an additional dose of naproxen placebo tablets.
  - For each subject, the data for up through Week 16 will be fixed prior to the Week 20 visit, and the fixed data will be prepared.
- 3) The blind will be maintained, including for the study sponsor, until the key code is opened after the data have been fixed for all subjects in Week 24. In addition, in order to eliminate any bias that could affect the study assessments, to the extent possible, the blind will be maintained with respect to the study site and the subject even after the opening of the study sponsor key code.

#### 3.2. Schedule of Study Procedures

#### 3.2.1. Test/Observation Schedule

Statistical Analysis Plan Protocol No. MT-5547-J01

Mitsubishi Tanabe Pharma Corporation (1) Test/Observation Schedule from informed consent to Week 48 of treatment period (if a joint replacement procedure is not going to be performed)

| | ľ | | | | | | Treatm | Treatment period | | | | | | | | Treatment period | eriod | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Тојиј | Screening | Pre-treatment<br>of observation<br>neriod | Day1<br>Baseline | Week1 | Week2 | Week4 | | Week12 | Week16 | Week 20 | Week 24 | Week 28 | Week 32 | Week 36 | Week 40 | 4 | Week 48 | At<br>withdrawa |
| Visit times (visit window) | consen<br>t | Day -37 | Day -7 ~-1<br>(±3) | | Day 8 | Day 15<br>(±3) | Day 29<br>(#7) | Day 57<br>(#1) | Day 85 | Day 113 | Day 141 | Day 169<br>(#7) | Day 197<br>(±7) | Day 225<br>(±7) | Day 253<br>(±7) | Day 281<br>(#7) | Day 309<br>(47) | Day 3.37<br>(#7) | |
| Visit Number | | - | 7 | 3 | 4 | \$ | Н | 7 | Н | - | - | 11 | - | - | + | $\vdash$ | + | 17 | |
| Written informed consent | × | | | | | | | | - | | | | | | | | | H | |
| Eligibility confirmed | | × | х | × | | | | | 1 | 1 | 1 | 1 | | 1 | | | | 1 | T |
| Demographics | | × | | × | 1 | 1 | 1 | | | | | | | | 1 | 1 | 1 | 1 | 7 |
| Randomir ation | | | | × | T | 1 | 1 | 1, | , | , | , | , | , | , | , | , | , | | |
| Study drug SC administration | 1 | | | × | | 1 | <del> </del> | 4 | < | × | ۲ | ٧ | V | 4 | v | V | v | 1 | |
| Administration of naproxen | 1 | | | | Ť | Ī | † | $\dagger$ | † | | ļ, | ļ, | Ħ, | ļ | ļ | ļ, | , | | |
| Delivery of haproxen | İ | | | | Ì | | † | $\dagger$ | T | + | { × | \<br>\ | ٠× | < × | <× | < × | < × | × | × |
| Delignment of accountments on | 1 | | * | <b>*</b> | Ì | × | × | × | × | × | × | × | × | : × | × | × | × | | |
| Return of acetaminophen/check of | | | | × | | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| amount taken | I | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| [Efficacy] | | | | | | | | | | | | | | 1 | | | | | |
| NDS (commend of the north) | Ľ | | × | \<br>\<br>\ | | | $\parallel$ | | T | <b>↑</b> | Γ | | | | | | | | |
| WOMA C | İ | × | | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| PGA of OA | | × | | × | × | × | × | × | × | x | × | × | × | x | x | × | x | × | × |
| SF36 | | | | × | | _ | х | х | | x | | x | | x | | × | | × | × |
| EQ-5D-5L | | | | х | | | х | x | | х | | х | | × | | × | | × | × |
| [Safety] | | | | | | | | | | | | | | | | | | | |
| Body weight (height: only at screening) | | × | | | | | | | | × | | | | | | | | × | × |
| Vital cions | | × | | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| ROG | | × | | | | | | - | | | | | | | | | | x | × |
| Physical examination | | × | | | | | | | | Н | | × | | × | | | | × | × |
| Orthostatic blood pressure | | x | × | × | | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Injection site assessment | | | | × | | | × | × | × | × | × | × | × | × | × | × | × | | |
| Joint Pain Questionnaire | | × | | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Autonomic Nerve Questionnaire | | × | | × | | | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Neurological evaluation | | × | | X<br>(brief | | X<br>(brief | u 2 | <b>~</b> 2 | <u>.</u> a | <u> </u> | (brief | X<br>(brief | (Brief | X<br>(brief | version) | (brief | (brief | × | × |
| Radiology (bilateral knees, hlps. | | × | | | | | ⊢ | - | - | ⊢ | | | | | | | | × | × |
| Shoulders) MRI testing | | | | | | | | | | | | | l | | | | | | |
| (evaluated joint, contralateral joint, | | × | | | | | | | | | | | | | | | | | |
| MRI testing (joint of joint replacement | | | | | | | T | | | | | | | | | T | | | × |
| Surgery ) | ľ | | | - | | I | | | İ | | | | | | | | | 1 | × |
| At ioint nain worsening | | | | | Ţ, | | | | | T | | ľ | | ľ | | Ī | T | , | |
| (Imaging [X-ray, MRI] assessments) | | | | | | П | Ħ | | | | | | | | | | | î | × |
| JOA Score | | | | | | | | | | | | | | | | | | | × |
| Laboratory testing | | × | | × | | 1 | × | × | × | × | 1 | × | 1 | × | | × | | × | × |
| Pregnancy test (for WOCBP)11 | | × | | × | | | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Bone density <sup>12</sup> | | × | | | | | 1 | 1 | 1 | 1 | | 1 | | 1 | | 1 | T | × | × |
| Urinalysis | | × | | × | | | | 1 | | × | | × | | | 1 | | | × | × |
| [Pharmacoldinetics] | Į | | | , | | | | , | , | | ľ | , | ľ | , | | | , | | ], |
| PK measurements | | | | ,x | × | × | × | × | × | k i | | ž, | Ī | ķ | | ķ | ķ | <b>,</b> | <b>*</b> |
| ADA antibody | | | | ž | | | | | | × | | × | | | | 1 | | 4 | 1 |
| lower | | | | | | | F | | | | | - | | | Ī | | | | ļ |
| | I | | | | | T | ┼<br>¶ | T | T | ┼<br><b>\</b> | Γ | <b>┬</b> | П | <u>Γ</u> | Γ | Γ | Ħ | | |


(2) Test/Observation Schedule of post-treatment observation period (if a joint replacement procedure is not going to be performed)

| | Pe | st-treatmen | t observati | on period ( | 20 weeks) <sup>14</sup> | At |
|---|---|---|---|---|---|---|
| | Week 52 | Week 56 | Week 60 | Week 64 | Week 68 | At<br>withdra<br>wal |
| Visit times (visit window) | Day 365<br>(±7) | Day 393<br>(±7) | Day 421<br>(±7) | Day 449<br>(±7) | Day 477<br>(±7) | |
| Visit Number | 18 | 19 | 20 | 21 | 22 | |
| Written informed consent | | | | | | |
| Eligibility confirmed | | | | | | |
| Demographics | | | | | | |
| Randomization <sup>1</sup> | | | | | | |
| Study drug SC administration <sup>2</sup> | | | | | | |
| Administration of naproxen | | | | | | |
| Delivery of naproxen | | | - | | | |
| Return of naproxen | | | | | | |
| Delivery of acetaminophen | | | | | <u> </u> | |
| Return of acetaminophen/check of amount taken <sup>3</sup> | | | | | | |
| amount taken Concomitant medications | x | X | x | х | X | X |
| [Efficacy] | 1 -12 | | | | 1 | |
| NRS (average daily pain) <sup>4</sup> | | | | | | |
| WOMAC <sup>5</sup> | Х | | x | | х | X |
| PGA of OA | X | | X | | х | X |
| SF-36 | | | | | х | X |
| EQ-5D-5L | <u> </u> | | · - | | x | X |
| [Safety] | | | • | | | |
| Body weight (height: only at screening) | | | | | x | x |
| Vital signs <sup>6</sup> | X | | | | X | X |
| ECG | | | | | | |
| Physical examination | | | | | X | X |
| Orthostatic blood pressure | X | | | | X | X |
| Injection site assessment | ! | | | | | |
| (30 minutes after administration) | x | | | | x | X |
| Joint Pain Questionnaire Autonomic Nerve Questionnaire | X | | | | X | X |
| Neurological evaluation | X<br>(brief<br>version) | | - | | X | X |
| Radiology (bilateral knees, hips, | | | | | | ** |
| shoulders) <sup>7</sup> | | | | | X | X |
| MRI testing<br>(evaluated joint, contralateral joint,<br>knee or hip joints with K-L≥3) <sup>7</sup> | | | | | | |
| MRI testing (joint of joint replacement surgery) | | | · | | | X |
| Adverse events | <del></del> | | | | <b>→</b> | X |
| At joint pain worsening | <del></del> | | | | <b>├</b> | x |
| (imaging [X-ray, MRI] assessments) <sup>8</sup> | ļ . | | | - | | ļ <u>.</u> |
| JOA Score <sup>9</sup> | | | - | - | <del> </del> | X |
| Laboratory testing | | | | | X | X |
| Pregnancy test (for WOCBP) <sup>11</sup> | X | | 1 | - | X | X |
| Bone density 12 | 1 | - | - | - | | |
| Urinalysis | | <u> </u> | | <u> </u> | X | X |
| [Pharmacokinetics] | | T | | | | T +, |
| PK measurements | X | X | | - | X | X |
| ADA antibody | | I | l | L | X | X |
| [Other] | <del> </del> | | · · | | | |

- Patients will be randomized (enrolled at the start of the treatment period) after all of the assessments through the pretreatment observation period have been completed.
- 2) Investigational drug or comparative drug will be administered subcutaneously after all of the safety assessments, efficacy assessments, and collection of blood samples for pharmacokinetic assessments have been completed, and patients will be kept under supervision at the study site for 30 minutes after the administration of the study drug or comparative drug.
- 3) The dose of acetaminophen taken will be checked based on the treatment diary. Every night, patients will record in their treatment diaries the amount (number of tablets) of acetaminophen they took that day.
- 4) Every night (and as a rule at the same time) from the start of the pre-treatment observation period until the day before Week 16, patients will use the IVRS to report the mean pain on walking for the previous 24 hours (NRS data). Patients will receive instruction in how to use the IVRS on the day of the visit at the start of the pre-treatment observation period.
- 5) The WOMAC score at screening will be assessed for the right knee joint, the left knee joint, the right hip joint, and the left hip joint, and the index joint will be determined based on the WOMAC pain subscale scores. At the other time points, the WOMAC score will be assessed for the index joint only.
- 6) If the pulse is less than 45 bpm at an assessment time point after investigational drug or comparative drug administration, electrocardiography will be performed and the patient carefully examined for cardiac function abnormalities.
- 7) Screening:

The following imaging tests will be performed for patients who meet the study eligibility criteria, and the images will be submitted to a central adjudication office. Imaging tests will also be performed if the central adjudication office requests that additional tests be conducted.

- · X- ray tests: Both knee joints, both hip joints, both shoulder joints
- · MRI tests: The index joint, the joint opposite the index joint, and any knee or hip joints with a K-L grade of 3 or more MRI tests will be performed as needed by the (sub) investigator.

A check will be performed by the day specified below to make sure that the results of the central assessments meet the study enrollment criteria.

- · X-ray tests: By the start of the pre-treatment observation period
- · MRI tests: By baseline

If the results of the central assessments cannot be confirmed by the specified day, then re-screening will be performed. After baseline:

At week 16, 48 (or at discontinuation of the treatment period) and at 68 weeks (or at the early discontinuation of the post-treatment observation period), images will be submitted to the central adjudication office. If the (sub) investigator determine that there is an abnormal finding compared to normal osteoarthritis, MRI tests will be performed as needed. The images will be submitted to a central adjudication office. Imaging tests will also be performed if the central adjudication office requests that additional tests be conducted, and the images submitted to the central adjudication office (for more detailed information, see in the text "9.2.4.1.11 Imaging Tests").

#### Week 16:

The X-ray tests (both knee joints, both hip joints, both shoulder joints) will be performed by the (sub) investigator. The images will be submitted to a central adjudication office. The (sub) investigator will check the X-ray images before administered the investigational drug or comparative drug to determine whether or not investigational drug or comparative drug should be administered. If any abnormalities are found, investigational drug or comparative drug administration will be postponed. If the central adjudication office rules out adjudicated arthropathy, investigational drug or comparative drug administration will be resumed.

At discontinuation of the treatment period and discontinuation of the post-treatment observation period

The X-ray tests (both knee joints, both hip joints, both shoulder joints) will be performed by the (sub) investigator. The images will be submitted to a central adjudication office. If more than 30 days have passed since the last images were taken, images will be taken again. If not more than 30 days have passed, imaging tests will be performed if the (sub) investigator determines that it is necessary.

- If joint replacement surgery is required, the MRI tests of the joint of surgery will be performed (for more detailed information, see in the text "9.2.4.1.13 Post-joint Replacement Procedure Assessment").
- 8) If a patient experiences a sudden worsening of pain that would not occur in the normal course of osteoarthritis, the (sub) investigator will postpone investigational drug or comparative drug administration, and perform imaging test (X-ray and MRI) of the affected joint. Imaging test (X-ray and MRI) of other joints will be performed as needed by the

13)

(sub) investigator. Imaging tests will also be performed if the central adjudication office requests that additional tests be conducted. All images will be submitted to the central adjudication office. The results of the central assessment will be checked by the (sub) investigator. The investigational drug or comparative drug administration will be postponed until the central adjudication office rules out adjudicated arthropathy. If adjudicated arthropathy is ruled out by the central assessment, then study treatment will be resumed. If the result of the central assessment is adjudicated arthropathy, then study treatment must be discontinued.

- 9) Assessments of the joint by JOA score at discontinuation will be performed for patients who required joint replacement surgery during the study.
- 10) Hematology and blood biochemistry tests will be performed. HbA1c, HBs antigen, HBs antibody, HCV antibody, and HIV antibody will be measured only at screening.
- 11) At screening, the pregnancy test will be performed using serum. At all other time points, the pregnancy test will be performed using urine. Furthermore, pregnancy tests will not be performed for postmenopausal females who have been amenorrheic for at least 1 year or for females who have undergone a surgical hysterectomy or bilateral ovariectomy. If a positive result is obtained on a urine pregnancy test, a serum pregnancy test will be performed. If a negative result is obtained on a serum pregnancy test, the study can be continued for the patient. If the serum pregnancy test is also positive, study treatment will be discontinued.
- 12) Bone density will be measured only at those study sites that are capable of performing measurements using the DEXA method. If it can not be measured at screening period, it may be measured during the pre-treatment observation period.
- 14) The Week 64 assessments may be performed by telephone.
- 15) The blood samples will be collected before the investigational drug or comparative drug is administered.
- 16) If a subject discontinues during the treatment period, a post-treatment observations will be performed at 4, 8, 12, 16, 20 and 24 weeks after the administration of the last dose of the investigational drug or control drug for the same parameters as those evaluated at the corresponding visits for completers. However, blood sample collection for pharmacokinetic evaluation is performed only 24 weeks after the last dose (blood sample collection for PK measurement is not necessary 4, 8 and 12 weeks after the last dose, which correspond to Weeks 48, 52 and 56 of the treatment period, respectively, for completers). The allowable time window for each evaluation time point is plus or minus 7 days.

The assessments at 12, and 20 weeks after the last dose administered to subjects discontinuing in the treatment period may be performed by telephone.

If the day of discontinuation from the treatment period and the day of discontinuation from the post-treatment observation period are the same (if the patient discontinued from the treatment period without proceeding to the post-treatment observation period), the assessments that are to be performed at discontinuation from the treatment period will be performed.

| Discontinuation<br>from the<br>treatment<br>period | 4 weeks<br>after the<br>last dose | 8 weeks<br>after the<br>last dose | 12 weeks<br>after the<br>last dose | 16 weeks<br>after the<br>last dose | 20 weeks<br>after the<br>last dose | 24 weeks<br>after the<br>last dose | Discontinuation<br>from the post-<br>treatment<br>observation period |
|---|---|---|---|---|---|---|---|
| Completed of the treatment period | Week 48 | Week 52 | Week 56 | Week 60 | Week 64 | Week 68 | Discontinuation<br>from the post-<br>treatment<br>observation period |

If the assessments at discontinuation are included in the allowable time window for each assessment time point, the parameters that are to be assessed at discontinuation will be assessed. Subsequently, at each time point after the last dose, the corresponding post-treatment assessments will be performed.

If not more than 30 days have passed since the last images were taken, imaging will not have to be performed again, but may be performed if the (sub) investigator determines that it is necessary. The tests at discontinuation and post-joint replacement procedure test/observation will be performed for patients who required joint replacement surgery during the study. Imaging test (X-ray and MRI) will be submitted to a central adjudication office (for more detailed information, see "9.1.1 (3) Post-joint replacement procedure test/observation schedule). If the assessments at discontinuation are not performed before the joint replacement procedure is performed, then images from before the procedure will be obtained and sent to the central adjudication office.

17) The screening period is from "the screening start date" to the day before "the pre-treatment observation period start date," and the screening start date and end date are defined to be consistent with the allowable time window of "the pre-

treatment observation period" (for example, if the pre-treatment observation period is 4 days, the maximum screening period is the 30 days from Day-34 to Day-5, and if the pre-treatment observation period is 10 days, the maximum screening period is the 30 days from Day-40 to Day-11).

At each study visit after the baseline date, the assessments that are performed by the patients themselves (WOMAC, PGA, joint pain questionnaire, SF-36, EQ-5D-5L, survey of autonomic symptoms) will be performed before all of the other assessments (including the assessments that are performed by the (sub) investigator) (except for cases where imaging tests are performed on a different day).

#### (3) Post-joint replacement procedure test/observation schedule

| | After surgery <sup>1</sup> | Long-term <sup>1</sup> |
|---|---|---|
| Follow-up day (visit window) | Follow-up survey, 4 weeks post-<br>operative | Follow-up survey 2, 20 weeks post-<br>operative |
| | 29 days post-operative (±5 days) | 141 days post-operative (±7 days) |
| Concomitant medications | X | X |
| [Safety] | | |
| Vital signs | X | X |
| Joint Pain Questionnaire | X | X |
| JOA score <sup>2</sup> | X | X |
| Radiology (bilateral knees, hips, shoulders) | X | X |
| Adverse events | <del></del> | <b>→</b> |
| At joint pain worsening (imaging [X-ray, MRI] assessments)3 | <del></del> | <b>→</b> |

- Information about the procedure, including prosthesis replacement and/or the extent of surgery wound healing, will be collected.
- 2) The condition of the joint following joint replacement surgery will be assessed using the JOA Score.
- 3) If a sudden worsening of pain that does not occur in the normal progression of osteoarthritis occurs, the (sub) investigator will perform imaging test (X-ray and MRI) of the affected joint. Imaging test (X-ray and MRI) of other joints will be performed as needed by the (sub) investigator. Imaging tests will also be performed if the central adjudication office requests that additional tests be conducted. All images will be submitted to the central adjudication office.

#### 3.3. Sample Size and Power Considerations

The original target sample size is 568 treated subjects (142 subjects per group)
(MT-5547 1 mg q4w group: 142 subjects; MT-5547 3 mg q4w group: 142 subjects; MT-5547
6 mg q8w group: 142 subjects; placebo group: 142 subjects)

After initiation of this study, based on the recommendations from the IDMC, the 3 mg q4w and 6 mg q8w groups were removed and 1 mg q8w group was newly added to the treatment groups.

The amended target sample size is 506 treated subjects, including the subjects who were randomized to 1 mg q4w/placebo groups before the amendment (approximately 40 subjects per group) and the subjects who are randomized to 1 mg q4w/1 mg q8w/placebo groups with the ratio of 1:1:1 after the amendment (142 subjects per group).

(MT-5547 1 mg q4w group: 182 subjects; MT-5547 1 mg q8w group: 142 subjects; placebo group: 182 subjects)

In addition, 57 patients each were enrolled in the MT-5547 3 mg q4w and 6 mg q8w groups prior to the protocol amendment (Ver. 04.00.00000) and were discontinued from study drug based on the recommendations from the IDMC. Thus, enrollment of 563 subjects is planned for this study in total.

#### The original rationale at the initiation of the study

Because this study is being conducted as a placebo-controlled study, in order to detect a statistical difference between the MT-5547 groups and the placebo group, the mean intergroup difference relative to placebo in both the change from baseline in the WOMAC pain subscale score and the change from baseline in the physical function subscale score at Week 16 for the MT-5547 3 mg SC q4w, 6 mg SC q8w, and 1 mg SC q4w groups was set at 1.1, and the standard deviation 2.5, on the basis of the results obtained in the overseas P2a study (R475-PN-0901) and the overseas P2b study (R475-PN-1227) (Table 3.3-1). The effect relative to placebo in the P3 study of 5 mg and 10 mg of tanezumab, another NGF inhibitor, was 0.81 to 1.21 in the WOMAC pain subscale score and 0.98 to 1.25<sup>24), 25)</sup> in the WOMAC physical function subscale score, and it therefore appears that a mean difference between the MT-5547 groups and placebo of 1.1 is a realistic assumption. It also appears that the minimum clinically significant difference in each WOMAC score will be around 0.67 to 0.75 <sup>26), 27)</sup>. The aforementioned intergroup difference of 1.1 exceeds the minimum clinically significant difference, and therefore seems to be an appropriate value to use for the intergroup difference. Based on a one-sided significance level of 2.5% and multiplicity adjustment based on a gate keeping method using a graphical approach, the power for MT-5547 3 mg SC q4w, 6 mg SC q8w, and 1 mg SC q4w will be 90%, 88%, and 88%, respectively, for the primary endpoint, and 82%, 79%, and 79%, respectively, for the key secondary endpoint. A 2-sample t-test will be used for the tests in each step. Based on this assumption, the number of subjects who will complete 16 weeks of treatment in each group will be 120.

Furthermore, because the proportion of missing data for the primary endpoint and the key secondary endpoint at Week 16 is around 15% according to Table 3.3-1, it is being assumed that the proportion of missing data at Week 16 will be 15%, and the number of patients per group is therefore being set at 142.

#### The rationale after the changes in treartment groups

Assuming the absolute treatment difference of 1.1 between the MT-5547 1 mg SC q8w groups and placebo in both the change from baseline in the WOMAC pain subscale score and

the change from baseline in the physical function subscale score at Week 16 with an associated standard deviation of 2.5 based on the original rationale at the initiation of the study, the number of patients per group after the protocol amendment (Ver. 04.00.00000) is planned to 142 subjects per group. The structure of statistical hypotheses have been changed due to the removal of 3 mg q4w / 6 mg q8w groups and the addition of 1 mg q8w. It is noted that approximately 40 subjects per group were randomized to 1 mg q4w / placebo groups before the amendment. For evaluation on 1 mg q4w, since subjects are randomized to 1 mg q4w / placebo at the same time with the same ratio of 1:1 regardless of pre- or post- amendment, analyses will be performed with pooled comparable data including pre- and post- amendment data on 1 mg q4w / placebo (1 mg q4w group: 182 subjects; placebo group: 182 subjects). For evaluation on 1 mg q8w, analyses will be performed with only the post-amendment data (1 mg q4w group: 142 subjects; 1 mg q8w group: 142 subjects; placebo group: 142 subjects). For four null hypotheses, based on multiplicity adjustment based on a gate keeping method using a graphical approach (Figure 8.2.1-1 in section 8.2.1 of SAP for database at week 16), the power for MT-5547 1 mg SC q4w and 1 mg SC q8w will be 97% and 92% for the primary endpoint, 94% and 87% for the key secondary endpoint, respectively.

Table 3.1-1 Change From Baseline at Week 16 in the WOMAC Pain and Physical Function Subscale Scores

| | | REGN St | udy R475 | -PN-1227 | 7 | REC | 3N Study | R475-PN | -0901 |
|---|---|---|---|---|---|---|---|---|---|
| | Placebo<br>(N=83) | MT-5547<br>1 mg<br>(N=85) | MT-5547<br>3 mg<br>(N=84) | MT-5547<br>6mg<br>(N=85) | MT-5547<br>9 mg<br>(N=84) | Placebo<br>(N=55) | MT-5547<br>0.03<br>mg/kg<br>(N=53) | MT-5547<br>0.1<br>mg/kg<br>(N=53) | MT-5547<br>0.3<br>mg/kg<br>(N=54) |
| | Ch | ange fron | n baseline | in WOM | IAC pain | subscale | score | | |
| Baseline | 6.43 | 6.33 | 6.35 | 6.10 | 6.53 | 5.9 | 5.7 | 6.1 | 6.4 |
| n <sup>1)</sup><br>Mean <sup>1)</sup><br>(SD) <sup>1)</sup> | 71<br>-2.43<br>(2.38) | 75<br>-3.49<br>(2.06) | 78<br>-3.39<br>(2.44) | 77<br>-3.07<br>(2.34) | 79<br>-3.81<br>(2.49) | 44<br>-2.4<br>(2.18) | 47<br>-2.7<br>(1.89) | 44<br>-3.4<br>(2.53) | 41<br>-3.2<br>(2.24) |
| LSM <sup>2)</sup> | -2.25 | -3.35 | -3.33 | -3.03 | -3.65 | _ | _ | - | - |
| Diff. vs. Pbo <sup>3)</sup> | - | -1.10 | -1.08 | -0.78 | -1.40 | - | -0.6 | -1.1 | -0.8 |
| P value | - | 0.0025 | 0.0029 | 0.0304 | 0.0001 | - | 0.1486 | 0.0090 | 0.0488 |
| | Change f | rom basel | ine in W | OMAC pl | nysical fu | nction sul | oscale sco | ore | |
| Baseline | 6.15 | 6.11 | 6.09 | 5.94 | 6.20 | 5.9 | 5.9 | 6.2 | 6.2 |

| $n^{1)}$ | 70 | 75 | 78 | 76 | 80 | 44 | 47 | 44 | 41 |
|---|---|---|---|---|---|---|---|---|---|
| Mean <sup>1)</sup> | -2.12 | -3.21 | -3.28 | -2.97 | -3.51 | -2.3 | -2.9 | -3.4 | -3.1 |
| (SD) <sup>1)</sup> | (2.26) | (2.23) | (2.29) | (2.45) | (2.50) | (2.30) | (1.78) | (2.28) | (2.18) |
| LSM <sup>2)</sup> | -1.98 | -3.08 | -3.27 | -3.03 | -3.41 | - | - | - | - |
| Diff. vs. Pbo <sup>3)</sup> | - | -1.10 | -1.29 | -1.06 | -1.43 | - | -0.8 | -1.1 | -0.9 |
| P value | - | 0.0019 | 0.0003 | 0.0029 | < 0.0001 | 1 | 0.0693 | 0.0071 | 0.0245 |

- 1) n: number of subjects at Week 16; mean: arithmetic mean at Week 16; SD: standard deviation at Week 16. However, in REGN Study R475-PN-1227, the n includes WOMAC data from after treatment discontinuation.
- 2) LSM: MMRM least squares mean
- 3) Diff. vs. Pbo: Difference for each group relative to the placebo group in the MMRM least squares mean

#### 4. PLANNED ANALYSIS

#### 4.1. Interim Analysis

A First-Step Analysis of the data was conducted using database in 24 week. No alpha adjustment is necessary, as the week 16 efficacy analysis is the final primary analysis for efficacy.

#### 4.2. Final Analysis

This SAP for 68 week will be finalized before database lock in 68 week. The analysis for week 68 will be conducted after database lock in 68 week.

#### 4.3. Independent Data Monitoring Board

An independent data monitoring board will periodically assess unblinded data, and will make recommendations to the study sponsor regarding the appropriateness of continuing the study and about the need for protocol amendments.

The independent data monitoring board will include independent statistical and medical experts. For more details, the overseas independent data monitoring committee procedures (DMC Charter) will be followed.

#### 5. ANALYSIS POPULATIONS

The analysis of efficacy will be performed in the full analysis set (FAS). The principal analysis set for efficacy will be the modified FAS (mFAS). The analysis of safety will be performed in the safety analysis set (SAF). The analysis of pharmacokinetics will be performed in the pharmacokinetic analysis set.

The analysis sets are defined below. For the contents of the data review meeting, refer to a separate materials.

#### (1) Efficacy analysis sets

1) Randomized subjects (RAND)

#### 2) FAS

The FAS will consist of all randomized subjects except for the following subjects.

- Subjects who have not received study drug even once
- Subjects with no WOMAC pain subscale score (the primary endpoint) at baseline
- Subjects with no WOMAC pain subscale score (the primary endpoint) at any time point after randomization

#### 3) Modified FAS (mFAS)

The mFAS will consist of the FAS, except for the following subjects.

- Subjects who are randomized to 3 mg q4w group
- Subjects who are randomized to 6 mg q8w group

#### (2) SAF

The SAF will consist of all randomized subjects except for the following subjects

- Subjects who did not receive study drug even once
- Subjects for whom absolutely no post-randomization safety data are available

#### (3) Self-injection analysis set(SIAS)

The self-injection analysis set will consist of the mFAS, except for the following subjects.

- Subjects who never performed self-injection

#### (4) Pharmacokinetic analysis set (PK)

The pharmacokinetic analysis set will consist of subjects who have received investigational drug at least once and who had at least one non-missing post-dose serum drug concentration data.

#### (5) Anti-drug antibody (ADA) analysis set (ADA)

The ADA analysis set will consist of all treated subjects who received investigational drug or comparative drug at least once and who had at least one non-missing post-dose ADA result.

#### (6) Neutralizing anti-drug antibody (NAb) analysis set (NAb)

The NAb population includes all treated patients who received any amount of study treatment (drug or placebo; Safety Analysis Set), and either tested negative for ADA or tested positive for ADA with at least one non-missing NAb result (either "NAb negative" or "NAb positive") following the first dose of study drug or placebo.

#### (7) Concentration-Response analysis set (CR)

The CR polulation other than CRP will include all patiens who received any study drug and who had at least one non-missing serum MT-5547 concentration following the first dose of study drug and at least one non-missing WOMAC pain subscale score, WOMAC physical function subscale score, alkaline phosphatase (ALP), or bone

specific alkaline phosphatase (BAP) value, as applicable for each C-R assessment. Placebo group patients who received any study treatment (i.e., placebo) and who had at least one non-missing WOMAC pain subscale score, WOMAC physical function subscale score, ALP or BAP value will also included as a reference for each C-R assessment other than CRP. For CRP, the CR polulation will include all patiens who received any study drug and who had at least one non-missing serum MT-5547 concentration following the first dose of study drug and at least one non-missing CRP value which measured by Latex method. The data after the discontinuation will be excluded in CR population. For CRP, Placebo group patients who received any study treatment (i.e., placebo) and who had at least one non-missing CRP value which measured by Latex method will also included as a reference.

#### 6. STATISTICAL CONSIDERATIONS

#### 6.1. Descriptive Statistics

#### (1) Non-PK related

Continuous data will be summarized descriptively using the number in the analysis set (N), the number of observations (n), mean, standard deviation (SD), median, minimum and maximum. Categorical data will be summarized using frequency counts and percentages. The denominator for the percentages will be the total number of subjects in the treatment group and analysis population being presented, unless otherwise specified.

#### (2) PK related

Serum concentrations will be summarized descriptively using N, n, mean, SD, median, Q1, Q3, minimum and maximum by clinical study day (as defined in the protocol) and treatment group.

#### 6.2. Statistical Tests

All formal statistical tests of treatment effects will not be done. Point estimates will be accompanied with two-sided 95% CIs where applicable.

#### 7. DATA CONVENTIONS

#### 7.1. Analysis Variable Definitions

#### 7.1.1. Study Subjects

#### 7.1.1.1. Demographic and Other Baseline Characteristics

#### (1) BMI

BMI will be recalculated using the formula below and reported to 1dp.

BMI  $(kg/m^2)$  = weight at screening (kg) / {height at screening (m)}<sup>2</sup>

(2) Age(years)
If (month of date of consent > month of date of birth) or (month of date of consent = month of date of birth and day of date of consent >= day of date of birth), then Age (years) = year of date of consent - year of date of birth

if else case, then Age (years) = year of date of consent - year of date of birth -1.

#### (3) Time since osteoarthritis diagnosis (years)

Time since osteoarthritis diagnosis will be calculated using the formula below and reported to 1dp.

If (month of date of consent > month of osteoarthritis diagnosis) or (month of date of consent = month of date osteoarthritis diagnosis, and day of date of consent >= day of date of osteoarthritis diagnosis), then Time since osteoarthritis diagnosis (years) = (date of consent - date of osteoarthritis diagnosis) / 365.25\*

if else case, then Time since osteoarthritis diagnosis (years) = (date of consent – date osteoarthritis diagnosis -1) / 365.25\*.

Impute date of osteoarthritis diagnosis as the earliest possible date (i.e. first day of month if day is unknown or 1st January if day and month are unknown).

#### (4) Renal function (stage 1, stage 2, stage 3, stage 4, stage 5)

The stages of renal function are defined by the FDA guidance as follows<sup>[1]</sup>

| Stage | Description <sup>b</sup> | eGFR <sup>c</sup> |
|-------|--------------------------|---------------------|
| | | $(mL/min/1.73m^2)$ |
| 1 | Control (normal) | ≥ 90 |
| | GFR | |
| 2 | Mild decrease in | 60-89 |
| | GFR | |
| 3 | Moderate decrease | 30-59 |
| | in GFR | |
| 4 | Severe decrease in | 15-29 |
| | GFR | |
| 5 | End Stage Renal | <15 not on dialysis |
| | Disease (ESRD) | Requiring dialysis |

#### 7.1.1.2. Medical History

Medical history will be coded according to the MedDRA version 20.1.

<sup>\*1</sup> year = 365.25 days

#### 7.1.1.3. Prior or Concomitant Medication

Medications will be coded according to the WHO Drug Dictionary (WHO-DD) Sep 2017 B3 version.

(1) Prior Medication

Prior medications are defined as medications starting prior to the first dose of study drug.

(2) Concomitant Medication

Medications that are on-going or start after the first intake of study drug are classified as "Concomitant".

Assessment period is defined as the time from first dose of investigational product up to 28 days after the last dose of investigational product.

(3) Post-treatment Medication

Medications that are start after on-treatment period are classified as "Post-treatment Medication".

# 7.1.1.4. Treatment Duration, Treatment and Post-Treatment Observation Duration and Compliance

- (1) Treatment Duration
- 1) Treatment duration (days) = The date of last study drug injection the date of the first study drug injection + 28.
- 2) Criteria for pre-defined limit

Treatment duration period  $\ge 1$  day,  $\ge 29$  days,  $\ge 57$  days,  $\ge 85$  days,  $\ge 113$  days,  $\ge 141$  days, > 169 days, > 197 days, > 225 days,  $\ge 253$  days,  $\ge 281$  days and  $\ge 309$  days

- (2) Treatment and Post-Treatment Observation Duration
- 1) Treatment and Post-Treatment Observation duration (days) = Date of last study visit [up to end of the post treatment observation period] date of first study drug dose).
- 2) Criteria for pre-defined limit

Treatment and Post-Treatment Observation duration period  $\geq 1$  day,  $\geq 29$  days,  $\geq 57$  days,  $\geq 85$  days,  $\geq 113$  days,  $\geq 141$  days and  $\geq 169$  days,  $\geq 197$  days,  $\geq 225$  days,  $\geq 253$  days,  $\geq 281$  days,  $\geq 309$  days,  $\geq 337$  days,  $\geq 365$  days,  $\geq 393$  days,  $\geq 421$  days and  $\geq 449$  days

- (3) Treatment Compliance
- 1) Treatment compliance will be calculated using the formula below and reported to 1dp.

#### MT-5547

Treatment compliance(%) = (Number of injections of study drug during exposure period) / (Number of planned injections of study drug during exposure period on or before the time that the subject discontinues from the study)  $\times 100\%$ 

#### **Naproxen**

Treatment compliance(%) = (Number of adherence of naproxen during exposure period) /

(Number of planned adherence of naproxen during exposure period on or before the time that the subject discontinues from the study) x 100%

#### 2) Criteria for pre-defined limit

#### MT-5547

the number of injections of study drug: 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 the number of self-injection of study drug: 1, 2, 3, 4, 5 and 6

#### 7.1.2. Efficacy assessments

#### 7.1.2.1. WOMAC pain subscale score

WOMAC pain subscale score

$$= \frac{\text{sum of items from Section A 1 to Section A5 in questionnaire}}{5}$$

#### 7.1.2.2. WOMAC physical function subscale score

WOMAC physical function subscale score

$$= \frac{\text{sum of items from Section C 8 to Section C24 in questionnaire}}{17}$$

#### 7.1.2.3. WOMAC stiffness subscale score

WOMAC stiffness subscale score = 
$$\frac{\text{Section B 6 + Section B7 in questionnaire}}{2}$$

#### 7.1.2.4. WOMAC total score

WOMAC total score = 
$$\frac{\text{sum of items from Section A1 to Section C24 in questionnaire}}{24}$$

#### 7.1.2.5. SF-36 / EQ-5D-5L

• SF-36

Physical, Mental and Role social component summary will be calculated considering factor coefficients based on the 1995 Japan National Survey. The derivation of 8 subscales and three component is detailed in appendix 1.

• EQ-5D-5L

Utility Index Score will be calculated using the formula and Table below.[1]

Utility Index Score

- = 1 + [Estimation of the constant term(if all answer is not 1)]
- + [Sum of "estimation of coefficients corresponding to answer other than 1"]

| Item | Level | Estimation | Standard Error | P-value |
|-----------|-------|------------|----------------|----------|
| Intercept | | -0.060924 | 0.013625 | < 0.0001 |
| | 2 | - 0.063865 | 0.008996 | < 0.0001 |
| Mo | 3 | -0.112618 | 0.009287 | < 0.0001 |
| IVIO | 4 | -0.179043 | 0.010231 | < 0.0001 |
| | 5 | -0.242916 | 0.009425 | < 0.0001 |
| | 2 | -0.043632 | 0.008931 | < 0.0001 |
| Sa. | 3 | -0.076660 | 0.009972 | < 0.0001 |
| Sc | 4 | -0.124265 | 0.010129 | < 0.0001 |
| | 5 | -0.159659 | 0.008924 | < 0.0001 |
| | 2 | -0.050407 | 0.009205 | < 0.0001 |
| Ua | 3 | -0.091131 | 0.010005 | < 0.0001 |
| ua | 4 | -0.147929 | 0.009744 | < 0.0001 |
| | 5 | -0.174786 | 0.009115 | < 0.0001 |
| | 2 | - 0.044545 | 0.008354 | < 0.0001 |
| n.i | 3 | -0.068178 | 0.010052 | < 0.0001 |
| Pd | 4 | -0.131436 | 0.008985 | < 0.0001 |
| | 5 | -0.191203 | 0.009604 | < 0.0001 |
| | 2 | -0.071779 | 0.009701 | < 0.0001 |
| ٨٨ | 3 | -0.110496 | 0.010863 | < 0.0001 |
| Ad | 4 | -0.168171 | 0.009850 | < 0.0001 |
| | 5 | -0.195961 | 0.009164 | < 0.0001 |

Mo: mobility, Sc: self-care, Ua: usual activities, Pd: pain/discomfort, Ad: anxiety/depression

e.g ) If answer is [1 1 1 1 1], Utility Index Score is = 1 + 0 + 0 = 1. If answer is [1 1 3 2 1], Utility Index Score is = 1 + (-0.060924) + (-0.091131 - 0.044545) = 0.8034.

# 7.1.2.6. Response rate based on the OMERACT-OARSI criteria



Note that the criteria in the diagram above are based on standardized score between 0 and 100. For this study, WOMAC pain and physical function subscale score are between 0 and 10, so the absolute change required for response is the required change in the diagram above divided by 10; PGA is 1, 2, 3, 4 or 5, so the absolute change required for response is at least 1 point.

#### 7.1.2.7. Rescue Medication

Baseline amount of rescue medication is defined as the average of the non-missing values during 7 days prior to taking study drug. For each week, the average of the non-missing values between date collected WOMAC and next date collected WOMAC will be used.

#### 7.1.3. Safety Assessments

The on-treatment period is defined as the time from first dose of investigational product up to 28 days after the last dose of investigational product.

The post-treatment period is defined as the time after the on-treatment period to the end of the post treatment observation period or early termination date.

#### 7.1.3.1. Adverse Events

Adverse events will be coded according to the MedDRA version 20.1

(1) Treatment Emergent Adverse Events/ Treatment Emergent Serious Adverse Events (TEAEs/TESAEs)

An AE/SAE is classified as treatment emergent if it newly occurred after the first dose of study drug or if a pre-dose event increases in severity following the first dose of study drug during on-treatment period.

(2) Post-Treatment Adverse Events/ Treatment Serious Adverse Events

An AE/SAE is classified as post-treatment if it newly occurred after the on-treatment period or if the event after the on-treatment period increases in severity.

(3) Adverse Drug Reaction

A TEAE is considered "adverse drug reaction" if it has been assessed as having a "reasonable possibility" in relationship to the study drug.

(4) Adverse Event of Special Interest(AESI)

Adjudicated arthropathy(AA), sympathetic nervous system dysfunction, altered peripheral sensation, destructive arthropathy(DA) are defined as adverse events of special interest (AESI) for the sake of investigating the safety profile of MT-5547.

(5) Identified and Potential Adverse Events

Following are defined as identified and potential adverse event for the sake of investigating the safety profile of MT-5547.

- · Arthralgia related event
  - (PT) Arthralgia
  - (PT) Osteoarthritis
  - (PT) Arthritis
  - (PT) Joint stiffness
  - (PT) Joint swelling
  - (PT) Joint effusion
  - (PT) Synovitis
- Bone fractures related event

Any PT containing "fracture" but excluding Tooth Fracture and Subchondral Insufficiency fracture (that have been identified to be AAs)

- Joint swelling related event
  - (PT) Joint Swelling
  - (PT) Joint Effusion
- Altered peripheral sensation related event
  - (HLGT) Peripheral Neuropathies
  - (HLT) Paraesthsias and dysaesthesias
  - (HLT) Sensory abnormalities NEC
  - (PT) Myalgia
  - (PT) Hyperreflexia
  - (PT) Hyporeflexia
  - (PT) Areflexia

- Sympathetic nervous system dysfunction related event
  - (HLT) Autonomic nervous system disorders
  - (HLT) Cardiac conduction disorders
  - (PT) Syncope
- Hypersensitivity / anaphylaxis related event
  - (SMQ) Angioedema
  - (SMQ) Anaphylactic reaction
  - (SMQ) Hypersensitivity
  - (PT) Erythema
  - (PT) Prurigo
  - (PT) Pruritus
  - (PT) Pruritus Generalised
  - (PT) Rash Papular
- (6) Duration of Adverse Events

Duration of Adverse Events (days) = AE stop date – AE start date + 1

(7) Incidence Rate (per 100 patient-years)

For patients with events, number of patient years is calculated up to the date of the first event and for patients without event, it corresponds to the length of the study observation period. Incidence Rate will be calculated using the formula.

Incidence Rate = the number of patients with event  $\times$  100 / sum of observation periods for all patients (days)  $\times$  365.25\*

\* 1 year = 365.25 days

#### 7.1.3.2. Laboratory Tests

Listing of reference value in each laboratory parameters is detailed in appendix 3

(1) The Estimated Glomerular Filtration Rate (eGFR)

eGFR will be calculated as follows and reported to 1 dp.

eGFR =  $141 \times \min(S_{Cr}/\kappa, 1)^{\alpha} \times \max(S_{Cr}/\kappa, 1)^{-1.209} \times 0.993^{Age} \times 1.018$  [if female] × 1.159 [if Black]

 $S_{Cr}$  (standardized serum creatinine) = mg/dL

 $\kappa = 0.7$  (females) or 0.9 (males)

 $\alpha = -0.329$  (females) or -0.411 (males)

min = indicates the minimum of  $S_{Cr}/\kappa$  or 1

max = indicates the maximum of  $S_{Cr}/\kappa$  or 1

Age = years

- (2) Laboratory values below the limit of quantification
- 1/2 LLOQ (lower limit of quantification) will be used for BLQ (below the limit of quantification) data in summary statistics. ULOQ (upper limit of quantification) will be used for over the limit of quantification data in summary statistics.
- (3) Criteria for pre-defined

Potentially clinically significant values (PCSV) ranges will be applied to the laboratory test values as applicable (see Appendix 2 for PCSV definitions).

#### 7.1.3.3. Vital Signs

(1) Criteria for pre-defined

Potentially clinically significant values (PCSV) ranges will be applied to the vital sign parameter values as applicable (see Appendix 2 for PCSV definitions).

#### 7.1.3.4. ECG

(1) Criteria for pre-defined

Potentially clinically significant values (PCSV) ranges will be applied to the ECG parameter values as applicable (see Appendix 2 for PCSV definitions).

(2) QTcF

QTcF will be calculated as follows and reported to 1 dp.

 $QTcF (msec) = QT/RR^{1/3}$ 

RR = 60/HR

#### 7.1.4. Pharmacokinetics Evaluation

#### 7.1.4.1. MT-5547 Concentrations in Serum

For the calculation of the summary statistics, concentration values reported as below the limit of quantification (BLQ) will be set to 0. In the log-scaled figures, concentrations below the LLOQ imputed as LLOQ/2. The lower limit of quantification (LLOQ) is 7.8 ng/mL in neat human serum.

#### 7.1.4.2. Anti-Drug Antibodies in Serum

Anti-drug antibody variables will include ADA status (positive or negative) and titer as follows:

- Total subjects negative in the ADA assay analyzed at all time points
- · Pre-existing immunoreactivity a positive ADA response at baseline with all post-dose

ADA results negative, or a positive ADA response at baseline with all post-dose ADA responses less than 9-fold over baseline titer levels.

- Treatment emergent defined as any post-dose positive ADA response when baseline results are negative
  - ➤ Persistent A positive result in the ADA assay detected in 2 consecutive post baseline samples, separated by at least 16-week period [based on nominal sampling time], with no ADA-negative results in-between, regardless of any missing samples
  - ➤ Indeterminate A positive result in the ADA assay at the last collection time point analyzed only, regardless of any missing samples
  - > Transient Not persistent or indeterminate regardless of any missing samples
- Treatment boosted defined as any post-dose positive ADA response that is at least 9-fold over the baseline level when baseline is positive in the ADA assay
- · Titer Values
  - Titer category: low (titer <1,000); moderate  $(1,000 \le \text{titer} \le 10,000)$ ; high (titer >10,000)
- · Neutralizing ADA activity for samples positive in the ADA assay

#### 7.2. Analysis Visit Definitions

(1) Analysis visit definitions for efficacy endpoints and PK endpoints (MT-5547 Concentrations, ADA and Concentration-Response Relationships)

| Analysis visit | Nominal day | Window |
|----------------|-------------|-------------------------|
| Baseline | Day 1 | <day 1<="" td=""></day> |
| Week 1 | Day 8 | Day 2 to 11 |
| Week 2 | Day 15 | Day 12 to 21 |
| Week 4 | Day 29 | Day 22 to 43 |
| Week 8 | Day 57 | Day 44 to 71 |
| Week 12 | Day 85 | Day 72 to 99 |
| Week 16 | Day 113 | Day 100 to 127 |
| Week 20 | Day 141 | Day 128 to 155 |
| Week 24 | Day 169 | Day 156 to 183 |
| Week 28 | Day 197 | Day 184 to 211 |
| Week 32 | Day 225 | Day 212 to 239 |
| Week 36 | Day 253 | Day 240 to 267 |
| Week 40 | Day 281 | Day 268 to 295 |
| Week 44 | Day 309 | Day 296 to 323 |
| Week 48 | Day 337 | Day 324 to 351 |
| Week 52 | Day 365 | Day 352 to 379 |
| Week 56 | Day 393 | Day 380 to 407 |
| Week 60 | Day 421 | Day 408 to 435 |
| Week 64 | Day 449 | Day 436 to 463 |
| Week 68 | Day 477 | Day 464 to 491 |



# (3) For Radiology analysis visit definitions

| Analysis visit | Nominal day | Window |
|----------------|-------------|-------------------------|
| Baseline | Day 1 | <day 1<="" td=""></day> |
| Week 16 | Day 113 | Day 86 to 141 |
| Week 48 | Day 337 | Day 310 to 365 |
| Week 68 | Day 477 | Day 450 to 505 |

The date of the first dose of study drug is defined as Day 1.

Unless otherwise specified, baseline will be the last observed value of the parameter of interest prior to the first intake of study drug (this includes unscheduled visits). For other visits, if there

are multiple data in a window, the closest data to nominal day will be used. If the distance to the nominal day is the same, the data of later date will be used. For orthostatic blood pressure, if a retest is performed, the initial value is compared with the retest value, and the worst value is used.

#### 7.3. Data Handling Convention for Missing Data

(1) Non-PK related

Efficacy:

#### WOMAC

WOMAC scores will be computed when one pain, one stiffness, or 1-3 physical function items are missing. The missing items will be imputed by the mean of available items within the same subscale. The scores will be set to missing if more items are missing.

#### SF-36 / EO-5D-5L

- SF-36 subscale scores will be computed if at least 50% of items are available. The missing items will be imputed by the mean of available items.
- EQ-5D-5L index will be set to missing if any of the 5 dimensions is missing.

#### **Rescue Medication**

If there is no date collected WOMAC, nominal date will be used.

#### Safety:

#### Adverse events

If severity or relationship is found to be missing the most severe occurrence will be imputed for the summary of interest.

For AE start missing or partial dates, the AE will be treated as TEAE if it cannot be determined to be a non-TEAE.

#### Laboratery test

Regarding hyaline casts and epithelial cells, set "Null" for blanks(= not detected) with date data.

#### **Orthostatic Blood Pressure**

If a retest is performed, the initial value should be compared with the retest value, and the value with the worst value should be used.

#### Other safety:

For safety summaries, only observed data will be used. If a value is indeterminate or a reference

value because of a problem with a test sample, then this value will be handled as a missing value.

#### (2) PK related

For PK summaries, only observed data will be used. Missing PK data will not be imputed. The PK data handling will be confirmed during blinded data review (BDR). PK data that are considered "invalid" will be flagged in the listing. Due to the nature of PK data, some issues may only be discovered after PK data are unblinded. Should new issues identified post unblinding, and new data handling rules would have to be applied, a separate PK data handling document will be produced to provide detailed rationale and decision making. If there is clear evidence that PK sample handling errors or other factors identified after data unblinding and these errors have led to unexpected erroneous data, then these erroneous data will be regarded as "invalid", full explanations will be given in the PK data handling document.

#### 8. STATISTICAL METHODOLOGY

#### 8.1. Study Subjects

#### 8.1.1. Subject Disposition

Screened subject disposition will be summarized on the all subjects. Randmized subject disposition will be summarized by treatment group, combined MT-5547 and overall on the randomized population. Randomization details will be listed on the randomized population. Subject disposition will be listed on the randomized population.

#### 8.1.2. Analysis Populations

Analysis populations will be summarized by treatment group, combined MT-5547 and overall on the randomized population. Analysis populations will be listed on the randomized population.

#### 8.1.3. Site Enrollment

Investigator enrollment will be summarized by treatment group and overall on the randomized population.

#### 8.1.4. Demographic and Other Baseline Characteristics

The following demographic and other baseline characteristics will be used.

| | category | Descriptive |
|------------|--------------|-------------|
| Sex | Male, Female | |
| Age(years) | <65,>=65 | Yes |
| Height(cm) | | Yes |

| Weight(kg) | | Yes |
|---|---|---|
| BMI(kg/m2) | <25, >=25 and<30, >=30 | Yes |
| Race | Japanese, other | |
| Time since OA diagnosis (years) | <1, >=1 and <5, >=5 and <10, >=10 | Yes |
| Complication | Yes, No | |
| Index Joint | Knee, Hip | |
| K-L score | 1, 2, 3, 4 | |
| Renal function | stage 1, stage 2, stage 3, stage 4, stage 5 | |
| WOMAC pain | <6 | Yes |
| subscale score | >=6 | 103 |
| WOMAC Physical function subscale score | <6<br>>=6 | Yes |
| PGA | 1, 2, 3, 4, 5 | Yes |
| Pain site | Right Knee, Left Knee,<br>Right Hip, Left Hip,<br>Right Shoulder, Left<br>Shoulder | |
| Pretreatment drug | NSAIDs(Systemic use),<br>NSAIDs(Topical use),<br>Acetaminophen, Opioid,<br>Monoamine reuptake<br>inhibitor, Hyaluronic<br>acid, Pregabalin, Herbal<br>medicine, Other | |
| NSAIDs Inadequate<br>Pain Relief | Yes, No | |
| NSAIDs Intolerance | Yes, No | |
| Ever taken Opioid for Pain due to OA | Yes, No | |
| Opioid Inadequate<br>Pain Relief | Yes, No | |
| Opioid Intolerance | Yes, No | |
| Ever taken Acetaminophen for Pain due to OA | Yes, No | |
| Acetaminophen<br>Inadequate Pain Relief | Yes, No | |
| Acetaminophen Intolerance | Yes, No | |

| NSAID + Opioid + | |
|------------------------|---------|
| Acetaminophen | Yes, No |
| Inadequate Pain Relief | |

Demographic and other baseline characteristics will be summarized by treatment group, and before the protocol amendment and after the protocol amendment on the mFAS population. Demographic and other baseline characteristics will be summarized by treatment group, combined MT-5547 and overall on the FAS population. Demographic and other baseline characteristics will be listed on the randomized population.

#### 8.1.5. Medical History

Medical history will be summarized by treatment group, combined MT-5547 and overall on the FAS population. Medical history will be listed on the randomized population.

#### 8.1.6. Radiograph eligibility data

Radiograph eligibility data at pre-treatment will be summarized by treatment group, combined MT-5547 and overall on the FAS population. Radiograph data will be listed on the randomized population.

#### 8.1.7. Prior or Concomitant Medications

Prior medication used for OA and concomitant medication and post-treatment medication will be summarized separately by treatment group and combined MT-5547 on the FAS population. All prior and concomitant medication and concomitant therapy and post-treatment therapy will be listed on the randomized population.

# 8.1.8. Treatment Duration, Treatment and Post-Treatment Observation Duration and Compliance

Treatment duration and treatment and post-treatment observation duration will be summarized by treatment group and combined MT-5547 on the SAF population. Treatment compliance of MT-5547 and naproxen will be summarized by treatment group and combined MT-5547 on the FAS population. The number of MT-5547 self-injection will be summarized by the principal investigator or sub-investigator and the self-injections and by MT-5547 treatment group on the mFAS population. Treatment duration, treatment and post-treatment observation duration and compliance will be listed on the randomized population. Study drug interruptions will be listed on the randomized population.

#### 8.2. Efficacy Assessments

Efficacy assessment will be summarized by treatment group on the mFAS population.

#### 8.2.1. Other Efficacy Endpoints

WOMAC pain subscale score, WOMAC physical function subscale score, WOMAC

#### stiffness subscale score, WOMAC total score, WOMAC individual score and PGA

For the changes from baseline at each assessment time point in the WOMAC pain subscale score, the WOMAC physical function subscale score, the WOMAC stiffness subscale score, the WOMAC total score, WOMAC individual score and PGA, the analysis will be tested using the estimator of mixed effect model for repeated measurement (MMRM) approach. The model will include the treatment group, measurement time point, treatment group and measurement time point interaction, stratification factor K-L grade (2-3 or 4), and stratification factor evaluated joint (knee or hip) as factors, and the corresponding baseline and baseline and measurement time point interaction as covariates. The within-subject correlation structure will be unstructured, and the denominator degrees of freedom for the test statistics of estimated parameters will be approximated using the Kenward-Roger method. In case the model will not converge with the unstructured covariance structure, Heterogeneous Autoregressive (1) (ARH[1]), Heterogeneous Compound Symmetry (CSH), Autoregressive (1) (AR[1]) or Compound Symmetry(CS) covariance structure will be used instead in this order. MMRM that assumes that the missing mechanism is missing at random (MAR) is an analysis method in which missing values are not replaced. This model will be used to estimate the treatment effect in the mFAS when subjects continue receiving treatment through Week 68.

The sampel SAS code planned for the analysis is outlined below.



WOMAC score and PGA will be listed. In addition, change from baseline to week 68 in WOMAC pain subscale score, WOMAC physical function subscale score and PGA will be graphed by visit.

#### SF-36 / EQ-5D-5L

For the changes from baseline at each assessment time point in SF-36 eight subscale summary scores and three component summary scores / EQ-5D-5L visual analogue scale(VAS) and utility index scores, the same analysis method (MMRM) as above will be analyzed. SF-36 / EQ-5D-5L will be listed.

Proportions of subjects with improvement of 30%, 50%, 70% and 90% at each assessment time point compared to baseline in WOMAC pain subscale score, WOMAC physical function subscale score and improvement of 30%, 50% and 70% at each assessment time point compared to baseline in PGA

A generalized linear mixed-effects model (GLMM) by logit type for response variable will be used to evaluate these binary response variables. The denominator degrees of freedom for the test statistics of estimated parameters will be approximated using the Kenward-Roger method. The estimated response rate for each treatment group and placebo group and 95% confidence interval of the odds ratio of each of the MT-5547 1 mg q4w and MT-5547 1 mg q8w groups compared to the placebo group in each binary response variables will be calculated using this GLMM approach.

- The covariates: baseline and the interaction of baseline and measurement time point.
- The fixed factors: Treatment group, measurement time point, the interaction of treatment group and measurement time point, K-L grade (2-3 or 4), and evaluated joint location (knee or hip)
- Random factors: Measurement time point for subject specific with covariance structure of unstructured

The sample SAS code planned for the analysis is outlined below.



# Response rate based on the OMERACT-OARSI criteria at each assessment time point compared to baseline

Responder analyses for OMERACT-OARSI will be summarized at each assessment time point using the same GLMM approach in previous model.

#### Proportion subjects who used rescue medication

The proportion of subjects taking rescue medication in baseline and up to week 48 will be summarized by treatment group. The proportion of days on rescue medication use during treatment priod will be summarized at each week by treatment group. Number of average usage of rescue medication will be summarized at each week by treatment group.

#### 8.2.2. Assessment of self-injection

# Analysis with respect to a comparison of the doses administered by the principal investigator or sub-investigator up through Treatment Week 24 and the self-injections performed after Treatment Week 24

The doses administered by the principal investigator or sub-investigator up through Treatment Week 24 and the self-injections performed after Treatment Week 24 will be analyzed using the same method[Section 8.2.1] as for the WOMAC pain subscale score.

Theses analysis will be summarized based on the self-injection population.

#### 8.3. Safety Assessments

Safety assessments will be made on the SAF population.

#### 8.3.1. Adverse Events

Overall summary of TEAEs / Post-treatment AEs for the following will be conducted.

- Subjects with at least one AE
- Subjects with at least one adverse drug reaction
- Subjects with at least one SAE
- Subjects with at least one serious adverse drug reaction
- Subjects with at least one AESI
- Subjects with at least one severe AE
- Subjects with at least one AE leading to discontinuation of study drug
- Subjects with AE leading to death

The following summaries also will be conducted.

- TEAEs / Post-treatment AEs AEs by SOC and PT
- TEAEs / Post-treatment AEs related to drug reactions by SOC and PT
- TEAESI / Post-treatment AESI by SOC and PT
- TESAEs / Post-treatment SAEs by SOC and PT
- TESAEs related to drug reactions by SOC and PT
- TEAEs leading to discontinuation of study drug by SOC and PT

- TEAEs / Post-treatment AEs by SOC, PT and severity
- TEAEs related to drug reactions by SOC, PT and severity
- TEAEs by SOC, PT and relationship to study drug
- TESAEs by SOC, PT and relationship to study drug
- Identified TEAEs / Post-Treatment AEs by SMQ, HLGT, HLT and PT

Each of the summaries will be done by treatment group and combined MT-5547 at the subject level - multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum severity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility/no reasonable possibility) and/or the earliest duration.

The following will be listed.

- AE
- AESI
- AE leading to discontinuation of study drug
- SAE
- Death
- Joint replacements

#### adjudicated arthropathy

The number and percentage of patients with images requiring adjudicated arthropathy as well as the number and percentage of those patients with confirmed adjudicated arthropathy including all available follow-up data after baseline will be summarized by treatment group and combined MT-5547. Subtypes of AAs and outcomes of AAs will also be summarized. Time to event with AA will be analyzed using Kaplan-Meir approach and will be plotted by treatment group. Cox regression model will be used for descriptively comparing each treatment group to placebo by obtaining hazard ratio estimates along with 95% confidence intervals.

#### Incidence of AA will be summarized by treatment group and combined MT-5547.

Incidence rate ratio estimates and 2-sided 95% confidence interval will be computed using Generalized Estimating Equations with a log-linked Poisson model via the PROC GENMOD procedure if there are events in the placebo group. The model will specify the use of a Poisson probability distribution with an offset= log (patient-observation period days) and model terms for treatment-as-received and each randomization strata. If there is no event in the placebo group, incidence rate ratio will not be calculated and confidence intervals for the incidence rate difference will be computed using Wald method.

The incidence rate estimates for each arm, the estimates of the incidence rate ratio and incidence rate difference between MT-5547 and placebo will be summarized.

The SAS code planned for the analysis is outlined below.



#### Assessment of self-injection

- Analysis with respect to a comparison of the doses administered by the principal investigator or sub-investigator after treatment week 24 and the self-injections performed after treatment week 24

This analysis will be summarized using the data after treatment week 24 by the principal investigator or sub-investigator and the self-injections and by MT-5547 treatment group excluding MT-5547 3mg q4w and MT-5547 6mg q8w on SAF population.

Overall summary for the following will be conducted.

- Subjects with at least one TEAE
- Subjects with at least one adverse drug reaction
- Subjects with at least one TESAE
- Subjects with at least one serious adverse drug reaction
- Subjects with at least one AESI
- Subjects with at least one severe TEAE
- Subjects with at least one TEAE leading to discontinuation of study drug
- Subjects with TEAE leading to death
- Subjects with at least one abnormal NCS or CS for injection site assessment

The following summaries also will be conducted.

• TEAEs by SOC and PT

#### 8.3.2. Laboratory Tests

Absolute values and changes from baseline will be summarized at each assessment time point by treatment group for the following laboratory tests parameters.

| Laboratory Test Parameters | - | | | | <br> | <br> |
|---|---|---|---|---|---|---|
| | | Laboratory | Test | Parameters | | |

| Hematology | RBC, Hemoglobin, Hematocrit, MCHC, WBC, Platelet, Neutrophils, Lymphocytes, Monocytes, Basophils, Eosinophils |
|---|---|
| Biochemistry | AST, ALT, ALP, LDH, Gamma-GTP, Total protein, Albumin, Total cholesterol, Total bilirubin, BUN, Serum creatinine, eGFR, Na, K, Cl, Ca, HCO <sub>3</sub> -, Uric acid, Triglycerides, BAP, Inorganic phosphorus, CPK, CRP |
| Urinalysis | pH, Specific gravity, Creatinine, Phosphate<br>(Qualitative value): Glucose, Protein, Occult blood, Bilirubin,<br>Nitrite, WBC, Sendiment WBC, Hyaline casts, Epithelial cells,<br>Bacteria, Yeast, Ketones |

Shift table of clinically relevant categories will be presented for the following laboratory tests parameters.

All data will be listed.

#### 8.3.3. Vital Signs

Absolute values and changes from baseline will be summarized at each assessment time point by treatment group for the following parameters.

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate (bpm)
- Body Temperature(°C)

The percentage of subjects with vital signs pre-defined limit will be summarized. All data will be listed.

#### 8.3.3.1. Assessment of Orthostatic Blood Pressure with standing value minus supine value

Absolute values and changes from baseline will be summarized at each assessment time point by treatment group for the following parameters.

- Systolic blood pressure 1 minute after standing
- Diastolic blood pressure 1 minute after standing
- Pulse rate 1 minute after standing
- Systolic blood pressure 3 minute after standing
- Diastolic blood pressure 3 minute after standing
- Pulse rate 3 minute after standing

#### 8.3.4. ECGs

Absolute values and changes from baseline will be summarized at each assessment time point by treatment group for the following parameters.

Heart Rate (bpm)

- PR (msec)
- RR (msec)
- QRS (msec)
- QT (msec)
- QTcF (msec)

The percentage of subjects with ECG values outside pre-defined limit will be summarized. All data will be listed.

#### 8.3.5. Physical Examinations

Physical examination will be listed for the following parameters.

- General Appearance
- Neurological
- Eyes
- Ears, nose, throat
- Cardiovascular
- Respiratory
- Abdominal
- Hepatic
- Gastrointestinal
- Musculoskeletal
- Dermatological

#### 8.3.6. Bone density

Bone density will be summarized and listed for the following parameters.

- YAM(%) and T-score
- Femoral neck
- Total hip
- Lumber Vertebra

#### **8.3.7. JOA** score

JOA score will be listed. Spaghetti plots including all available follow-up data after baseline will be presented by treatment group and JR joint and the corresponding to joint.

#### 8.3.8. Radiograph

Adjudicated Arthropathy

Overall summary for adjudicated arthropathy will be conducted.

The following summaries for adjudicated arthropathy also will be conducted.

- Subtype of adjudicated arthropathy
- Subtype of adjudicated arthropathy meeting destructive arthropathy

- Incidence rate of adjudicated arthropathy
- Time to first event of adjudicated arthropathy

As regards time to first event adjudicated arthropathy, cox regression model will be used for descriptively comparing each treatment group to placebo by obtaining hazard ratio estimates along with 95% confidence intervals.

Each of the summaries will be done by treatment group and combined MT-5547.

All data will be listed.

#### Jonint Space Width

The following summaries for joint space width will be conducted.

- Non arthropathy adjucation joint with adjudicated arthropathy
- All joint with non adjudicated arthropathy subjects

Joint space width for AA will be summarized by treatment group and combined MT-5547. All data will be listed. Each of the summaries will be done by treatment group and combined MT-5547.

#### 8.3.9. Injection Site Assessments

Injection Site Assessments will be summarized at each assessment time point by treatment group. All data will be listed.

#### 8.3.10. Autonomic Symptoms Questionnaire

Absolute values and changes from baseline will be summarized at each assessment time point by treatment group for the following tests.

- total symptoms score
- total symptom impact scores

All data will be listed.

#### 8.3.11. Neurological Examinations

Neurological Examinations will be summarized by treatment group for the following tests.

- Cranial Nerve Exam
- Sensory Function
- Motor Function
- Reflexes
- Coordination

#### 8.3.12. Joint Pain Questionnaire

Joint pain questionnaire will be listed.

#### 8.3.13. Joint Replacement

Number and percentage of patients with joint replacement including all available follow-up data after baseline will be summarized by treatment group and combined MT-5547. Time to event with joint replacement including all available follow-up data after baseline will be analyzed using Kaplan-Meir approach and will be plotted by treatment group.

All data will be listed.

#### 8.4. Pharmacokinetics Evaluation

#### 8.4.1 Analysis of MT-5547 Concentration in Serum

Serum MT-5547 concentrations will be summarized at each nominal sampling point for each treatment group. All serum concentrations will also be listed.

Plots of the mean (+SD) concentrations (linear scales or log scales) will be presented by nominal time. Plots of the individual concentrations (linear scales or log scales) will be presented over actual sampling time. When the scale is linear, concentrations below the LLOQ are set to zero. In the log-scaled figures, concentrations below the LLOQ imputed as LLOQ/2.

#### 8.4.1. Analysis of Anti-Drug Antibody in Serum

Anti-MT-5547 antibody status and titers will be presented by nominal time.

The ADA variables described in Section 7.1.3.3 will be summarized using descriptive statistics by group/drug product in the ADA analysis set. Prevalence of pre-existing immunogenicity, treatment-emergent and treatment-boosted ADA will be assessed as absolute occurrence (N) and percent of patients (%), grouped by groups. For treatment emergent ADA, occurrence (N) and percent of patients (%) with persistent, transient and indeterminate ADA will be reported. The influence of treatment-emergent or treatment-boosted ADA assay response on individual PK profiles will be evaluated.

Listings of ADA status presented by subject, time point, and group will be provided.

Listings of ADA positivity and titers presented by subject, time point, and group will also be provided.

Correlation analysis of safety versus ADA and NAb positivity status may be performed on the SAF. Assessment will focus on the following safety events:

- Hypersensitivity (SMQ : Hypersensitivity [Narrow])
- Anaphylaxis (SMQ: Anaphylaxis[Narrow])

Number (%) of patients with the above mentioned safety events may be summarized by ADA positivity status, during the TEAE period.

In addition, correlation analysis of key efficacy endpoints versus ADA and NAb status may be summarized.

#### 8.4.2. Assessment of Concentration-Response Relationships

The scatter plot of each efficacy (WOMAC pain subscale score and WOMAC physical function subscale score) and safety variables (alkaline phosphatase, CRP and BAP value) vs. MT-5547 concentration at each time point by clinical study week will be presented for each dosing regimen, q4w (1 mg q4w and 3 mg q4w) and q8w (1 mg q8w and 6 mg q8w) and all dosing regimen (1 mg q8w, 1 mg q4w, 3 mg q4w and 6 mg q8w). Regarding the scatter plot of each efficacy (WOMAC pain subscale score and WOMAC physical function subscale score), the data after the discontinuation will be excluded. For safety variables, additional enlarged figures will be presented as needed.

In all plots, concentrations below the LLOQ were imputed to zero.

Additional analyses will be performed as necessary.

In accordance with the minutes of Blind Data Review Meeting conducted on 14<sup>th</sup> of Apr 2021 (BDRM), C-R analysis for CRP will include only the patients who have CRP values measured by Latex method throughout the study (Item No. 3 below).

| • | |
|---------------------------------------|--------------|
| Type | C-R analysis |
| Only measured as hsCRP | Not included |
| Baseline was measured as hsCRP, which | Not included |
| was changed to CRP during the study. | |
| Only measured as CRP | Included |



#### 9. DATA PRESENTATION CONVENTIONS

#### 9.1. Number of Digits to Report

#### (1) Non-PK related

| Statistic | Specification | Apply to |
|---|---|---|
| Minimum, Maximum | Same number of DPs as the data provided in the datasets | All original (i.e. non-derived) |
| | see section 7.3 | All derived data |
| Mean, Median, SD, SE,<br>Confidence intervals | One more DP than above | All |
| Percentages*1 | 1 DP | All |
| Ratios | 3 DPs | All |

Percentages: use 1 place beyond the decimal point, except for the following cases:

If the percentage is equal to 0, then leave blank, do not use (0)

\*

If the percentage is equal to 100, then use "(100)" without a decimal

# (2) PK and Concentration in Serum

| Statistic | Specification |
|------------------|--------------------------------------------|
| Individual value | 3 significant digits |
| Minimum, Maximum | Same number of DPs as the individual value |
| Mean, SD, Median | Same number of DPs as the individual value |

## 9.2. Treatments to Report

| Treatment | For TFLs |
|------------------------------------------|------------------|
| MT-5547 1 mg q8w | MT-5547 1 mg q8w |
| MT-5547 1 mg q4w | MT-5547 1 mg q4w |
| MT-5547 1 mg q4w and MT-5547 1 mg | MT-5547 Combined |
| q8w | |
| MT-5547 3 mg q4w | MT-5547 3 mg q4w |
| MT-5547 6 mg q8w | MT-5547 6 mg q8w |
| Placebo | Placebo |
| Placebo group and all active dose levels | Total |

# 9.3. Analysis Visits to Report

# (1) Non-PK related

# Efficacy:

| Analysis | Apply to | |
|----------|----------|-----------|
| Visit | | · · |
| | WOMAC | SF-36 and |
| | and PGA | EQ-5D-5L |
| Baseline | X | X |
| Week 1 | X | |
| Week 2 | X | |
| Week 4 | X | X |
| Week 8 | X | X |
| Week 12 | X | |
| Week 16 | X | X |
| Week 20 | X | |
| Week 24 | X | X |
| Week 28 | X | |
| Week 32 | X | X |
| Week 36 | X | |
| Week 40 | X | X |
| Week 44 | X | |
| Week 48 | X | X |
| Week 52 | X | |
| Week 56 | | |
| Week 60 | X | |
| Week 64 | | |

| Week 68 X X |
|-------------|
|-------------|

# Safety:

| Analysis Visit | Apply to | | | |
|---|---|---|---|---|
| | Laboratory<br>Tests | Injection Site<br>Assessments | Survey of Autonomic Symptoms | Vital Signs, Joint pain questionnaire |
| Baseline | X | X | X | X |
| Week 1 | | | | X |
| Week 2 | | | | X |
| Week 4 | X | X | X | X |
| Week 8 | X | X | X | X |
| Week 12 | X | X | X | X |
| Week 16 | X | X | X | X |
| Week 20 | | X | X | X |
| Week 24 | X | X | X | X |
| Week 28 | | X | X | X |
| Week 32 | X | X | X | X |
| Week 36 | | X | X | X |
| Week 40 | X | X | X | X |
| Week 44 | | X | X | X |
| Week 48 | X | | X | X |
| FU Week 4 | X | | X | X |
| FU Week 8 | | | X | X |
| FU Week 12 | | | | |
| FU Week 16 | | | | |
| FU Week 20 | | | | |
| FU Week 24 | X | | X | X |
| End of last | X | | | |
| observation | | | | |

| Analysis<br>Visit | Apply to | | | | |
|---|---|---|---|---|---|
| | ECGs, | Physical | Neurological | Radiograph | JOA |
| | Bone | Examinations* | Examinations, | | score** |
| | dencity* | | Orthostatic | | |
| | | | Hypotension | | |
| Baseline | X | X | X | X | |
| Week 1 | | | | | |
| Week 2 | | | X | | |
| Week 4 | | | X | | |
| Week 8 | | | X | | |
| Week 12 | | | X | | |
| Week 16 | | | X | X | |

| W71- 20 | [" | | V | |
|-------------|----|---|---|---|
| Week 20 | | | X | |
| Week 24 | | | X | |
| Week 28 | | | X | |
| Week 32 | | X | X | |
| Week 36 | | | X | |
| Week 40 | | | X | |
| Week 44 | | | X | |
| Week 48 | X | X | X | X |
| FU Week 4 | | | X | X |
| FU Week 8 | | | X | |
| FU Week 12 | | | | |
| FU Week 16 | | | | |
| FU Week 20 | | | | |
| FU Week 24 | | X | X | X |
| End of last | X | | | |
| observation | | | | |

Unscheduled visits, retests (same visit number assigned) and follow-up visits will not be displayed in by-visit summary tables, but will be included in the data listings.

#### (2) PK related

MT-5547 Concentrations, ADA and Concentration-Response Relationships for efficacy valiables (WOMAC pain subscale score and WOMAC physical function subscale score):

| Analysis | Apply to | : |
|----------|------------------------------------------|------|
| Visit | ) m 55.15 G | 1.54 |
| | MT-5547 Concentrations and | ADA |
| | Concentration-Response Relationships for | |
| | efficacy valiables (WOMAC) | |
| Baseline | X | X |
| Week 1 | X | |
| Week 2 | X | |
| Week 4 | X | |
| Week 8 | X | |
| Week 12 | X | |
| Week 16 | X | X |
| Week 24 | X | X |
| Week 32 | X | |
| Week 40 | X | |
| Week 44 | X | |
| Week 48 | X | X |
| Week 52 | X | |

<sup>\*</sup>Baseline is the screening assessment time point

<sup>\*\*</sup>Assessmets of the joint by JOA score at discontinuation will be performed for subjects who required joint replacement surgery during the study.

| Week 56 | X | |
|-----------|---|---|
| Week 68 | X | X |
| End of | | X |
| treatment | | |

Concentration-Response Relationships for safety valiables (ALP, CRP and BAP) and

| : | | |
|------------|------------------------------------|------|
| Analysis | Apply to | . "" |
| Visit | | |
| | Concentration-Response | |
| | Relationships for safety valiables | |
| | (ALP, CRP and BAP) | |
| Baseline | X | X |
| Week 1 | X | |
| Week 2 | X | |
| Week 4 | X | X |
| Week 8 | X | |
| Week 12 | X | |
| Week 16 | X | X |
| Week 24 | X | X |
| Week 32 | X | X |
| Week 40 | X | |
| Week 44 | X | |
| Week 48 | X | X |
| FU Week 4 | X | X |
| FU Week 8 | | |
| FU Week 12 | | |
| FU Week 16 | | |
| FU Week 20 | | |
| FU Week 24 | X | X |

#### 10. CHANGE FROM THE PROTOCOL

There are currently no changes to analysis from protocol.

#### 11. SOFTWARE

All statistical analyses will be performed using SAS version 9.3 or higher.

#### 12. REFERENCES

- [1] Shinya I, Takeru S, Ataru I, Shinichi N, Takashi F, et al. Developing a Japanese version of the EQ-5D-5L value set. J. Natl. Inst. Public Health.2015;64 (1): 47-55.
- [2] Fukuhara S, Suzukamo Y. Manual of SF-36v2 Japanese version: Institute for Health Outcomes & Process Evaluation research. Kyoto: 2004. Ver3/2011.

## **APPENDIX**

Appendix 1 SF-36v2 Scoring Algorithm<sup>[2]</sup>











Criteria for Potentially Clinically Significant Values (PCSV) Appendix 2

Mitsubishi Tanabe Pharma Corporation

| Parameter | PCSV | Comments |
|---|---|---|
| Clinical Chemistry | mistry | |
| ALT* | >3 and \le 5 ULN and baseline \le 3 ULN* >5 and \le 10 ULN and baseline \le 5 ULN >10 and \le 20 ULN and baseline \le 10 ULN >20 ULN | Enzyme activity must be expressed in ULN, not in IU/L. FDA DILI Guidance July 2009. Each category is calculated independently. * At least one level is required, multiple levels are optional for phase 2/3 studies. If it is desirable to get the distribution across the different PCSV levels, additional shift table on \$\leq 3, > 3\$ to \$\leq 5, > 5\$ to \$\leq 10\$, > 10 to \$\leq 20\$, and > 20 category for baseline vs. post baseline may be provided |

| Parameter | PCSV | Comments |
|---|---|---|
| AST* | >3 and $\leq$ 5 ULN and baseline $\leq$ 3 ULN* | Enzyme activity must be expressed in ULN, not in IU/L. |
| | $>$ 5 and $\leq$ 10 ULN and baseline $\leq$ 5 | FDA DILI Guidance July 2009. |
| | ULN $>10$ and $\leq 20$ ULN and baseline $\leq 10$ | Each category is calculated independently. |
| | ULN $>$ 20111 N and baseline $<$ 20111 N | * At least one level is required, |
| | | 2/3 studies. If it is desirable to get the |
| | | distribution across the different PCSV levels, additional shift table on |
| | | $\leq 3, > 3$ to $\leq 5, > 5$ to $\leq 10, > 10$ to $\leq 20,$ |
| | | and > 20 category tor baseline vs. post baseline may be provided |
| Alkaline<br>Phosphatase | >1.5 ULN and baseline $\leq$ 1.5 ULN | Enzyme activity must be expressed in ULN, not in IU/L. |
| | | FDA DILI Guidance July 2009. |


| Parameter | PCSV | Comments |
|---|---|---|
| Total Bilirubir | Total Bilirubin* >1.5 and $\leq$ 2 ULN and baseline $\leq$ 1.5 ULN* and baseline $\leq$ 2.0 ULN | Must be expressed in ULN, not in μmol/L or mg/L. Categories are cumulative. FDA DILI Guidance July 2009. |
| | | * At least one level is required, multiple levels are optional for phase 2/3 studies. If it is desirable to get the distribution of significant level, additional shift table on <1.5, >1.5 to <2.0 and > 2.0 category for baseline vs. post baseline may be provided |
| Conjugated<br>Bilirubin | (Direct Bilirubin >35% Total Bilirubin Conjugated bilirubin dosed on a case-and Total Bilirubin >1.5 ULN) and by-case basis. (Direct Bilirubin <=35% Total Bilirubin <=1.5 ULN) at baseline | Conjugated bilirubin dosed on a caseby-case basis. |

| Parameter | PCSV | Comments |
|---|---|---|
| ALT/AST and<br>Total Bilirubin | ALT/AST and (ALT >3 ULN and TBILI>2 ULN) and FDA DILI Guidance July 2009. Total Bilirubin baseline (ALT <=3 ULN or TBILI <=2 ULN) | FDA DILI Guidance July 2009. |
| | (AST >3 ULN and TBILI>2 ULN) and baseline (AST <=3 ULN or TBILI <=2 ULN) | |
| | (ALT >3 ULN and TBILI>1.5 ULN) and baseline (ALT <=3 ULN or TBILI <=1.5 ULN) | |
| | (AST >3 ULN and TBILI>1.5 ULN) and baseline (AST <=3 ULN or TBILI <=1.5 ULN) | |

(ALT >3 ULN and TBILI>2 ULN and FDA DILI Guidance July 2009. ALP < 2 ULN) and baseline (ALT <=3 ULN or TBILI <=2 ULN or ALP >=2 ALP < 2 ULN) and baseline (AST <=3 ULN or TBILI <=2 ULN or ALP >=2 (AST>3 ULN and TBILI>2 ULN and ULN) Total Bilirubin ALT/AST and and ALP

| Parameter | PCSV | Comments |
|---|---|---|
| CPK* | >3 and \le 10 ULN and baseline \le 3ULN* >10 ULN and baseline \le 10ULN | FDA Feb 2005. Am J Cardiol April 2006. Categories are cumulative. * At least one level is required, multiple levels are optional for phase 2/3 studies. If it is desirable to get the distribution of significant level, additional shift table on ≤3, >3 to ≤10, and > 10 category for baseline vs. post baseline may be provided |
| Creatinine | >150 µmol/L (Adults) and baseline < 150 µmol/L<br>>=30% change from baseline and <100% change from baseline<br>>100% change from baseline | Benichou C., 1994.<br>3 independent criteria |
| Uric Acid<br>Hyperuricemia<br>Hypouricemia | >408 µmol/L and <=408 µmol/L at baseline <120 µmol/L and >= 120 µmol/L at baseline | Harrison- Principles of internal Medicine 17 <sup>th</sup> Ed., 2008.<br>Two independent criteria |
| Blood Urea<br>Nitrogen | >17 mmol/L and <17 mmol/L at baseline | Two independent criteria |


Statistical Analysis Plan Protocol No. MT-5547-J01

| Parameter | PCSV | Comments |
|---|---|---|
| Chloride | | Two independent criteria |
| Hypochloremia | Hypochloremia <80 mmol/L and baseline ≥ 80 mmol/L | |
| Hyperchloremia | Hyperchloremia $>115$ mmol/L and baseline $\leq 115$ mmol/L | |
| Sodium | | Two independent criteria |
| Hyponatremia<br>Hypernatremia | <pre>&lt;129 mmol/L and baseline &gt; 129 mmol/L</pre> | |
| 16- | >160 mmol/L and baseline <160 mmol/L | |
| Potassium | | FDA Feb 2005. |
| Hypokalemia | $<3$ mmol/L and baseline $\geq 3$ mmol/L | Two independent criteria |
| Hyperkalemia | >5.5 mmol/L and baseline <5.5 mmol/L | |
| Total<br>Cholesterol | $\geq$ 7.74 mmol/L and < 7.74 mmol/L at baseline | Threshold for therapeutic intervention. |
| Triglycerides | >4.6 mmol/L and < 4.6 mmol/L at baseline | Threshold for therapeutic intervention. |

| Parameter | PCSV | Comments |
|---|---|---|
| Glucose<br>Hypoglycaemia<br>Hyperglycaemia | Glucose Hypoglycaemia (≤3.9 mmol/L and <lln) (="" and="">3.9 Hyperglycaemia mmol/L or &gt;=LLN) at baseline ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) and &lt; 11.1 mmol/L (unfasted); &lt;7 mmol/L (fasted) at baseline</lln)> | ADA May 2005.<br>ADA Jan 2008. |
| HbA1c | >8% and <= 8% at baseline | |
| Albumin | <25 g/L and >25 g/L at baseline | |
| CRP | >2 ULN or >10 mg/L (if ULN not provided) and <=2 ULN or <=10 mg/L (if ULN not provided) at baseline | FDA Sept 2005. |
| Hematology | | |
| WBC | <3.0 Giga/L and >=3.0 Giga/L at baseline (Non-Black); <2.0 Giga/L and >=2.0 Giga/L at | Increase in WBC: not relevant. |
| | baseline (Black)<br>≥16.0 Giga/L and < 16 Giga/L at baseline | To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L and <= 4.0 Giga/L at baseline | |

| Parameter | PCSV | Comments |
|---|---|---|
| Neutrophils | <pre>&lt;1.5 Giga/L and &gt;=1.5 Giga/L at baseline (Non-Black);</pre> | International Consensus meeting on drug-induced blood cytopenias, 1991. |
| | <1.0 Giga/L and >=1.0 Giga/L at baseline (Black) | FDA criteria. |
| Monocytes | >0.7 Giga/L <= 0.7 Giga/L at baseline | |
| Basophils | >0.1 Giga/L <= 0.1 Giga/L at baseline | |
| Eosinophils | (>0.5 Giga/L and >ULN) and (<=0.5 Giga/L or <= ULN at baseline) | Harrison- Principles of internal Medicine 17 <sup>th</sup> Ed., 2008. |
| Hemoglobin | ≤115 g/L and > 115 g/L at baseline for Three criteria are independent.<br>male; | Three criteria are independent. |
| | \( \frac{\geq 95 g/L}{2} \) at baseline for Female. | |
| | ≥185 g/L and <185 g/L at baseline for Male; | Criteria based upon decrease from baseline are more relevant than based on absolute value. Other categories |
| | $\geq$ 165 g/L and < 165 g/L at baseline for for decrease from baseline can be Female used ( $\geq$ 30 g/L, $\geq$ 40 g/L, $\geq$ 50 g/L). | for decrease from baseline can be used ( $\geq$ 30 g/L, $\geq$ 40 g/L, $\geq$ 50 g/L). |
| | Decrease from Baseline >20 g/L | |


| Parameter | PCSV | Comments |
|---|---|---|
| Hematocrit | ≤0.37 v/v and > 0.37 v/v at baseline for Male; ≤0.32 v/v and > 0.32 v/v at baseline forFemale | Two Criteria are independent |
| | $\geq 0.55$ v/v and $< 0.55$ v/v at baseline for Male; $\geq 0.5$ v/v and $< 0.5$ v/v at baseline for Female | |
| RBC | Female | Unless specifically required for |
| | $<$ 3 Tera/L and baseline $\geq$ 3 Tera/L | particular drug development, the |
| | ≥6 Tera/L and baseline < 6 | Otherwise, consider FDA criteria. |
| | Tera/L Male | |
| | <4 Tera/L and baseline ≥4 Tera/L | |
| | $\geq$ 7 Tera/L and baseline < 7 Tera/L | |
| Platelets | <100 Giga/L and >=100 Giga/L at baseline | International Consensus meeting on drug-induced blood cytopenias, 1991. |
| | ≥700 Giga/L and < 700 Giga/L at baseline | Two independent criteria |

| Parameter | PCSV | Comments | |
|---|---|---|---|
| Urinalysis | | | |
| Hd | <4.6 and > 4.6 at baseline | Two independent criteria | |
| | ≥8 and < 8 at baseline | | |
| Vital signs | | | |
| PR | ≤50 bpm and decrease from baseline ≥20 bpm | To be applied for all positions (including missing) except STANDING. | positions<br>except |
| | >120 bpm and increase from baseline>20 bpm | | |
| SBP | <ul> <li>Sommore and decrease from baseline (including missing singular)</li> <li>STANDING.</li> </ul> | all ) | positions |
| | ≥20 mmHg | | |
| DBP | <ul> <li>45 mmHg and decrease from baseline (including missing)</li> <li>10 mmHg STANDING.</li> </ul> | To be applied for all (including missing) STANDING. | positions<br>except |
| | >10 mmHg | | |


Statistical Analysis Plan Protocol No. MT-5547-J01


| Parameter | PCSV | Comments |
|---|---|---|
| Orthostatic Hypotension as per protocol, Orthostatic Hypotension confirmed by repeated assessment as per protocol | Su SBP < 160 mmHg - SBP St - Su $\le$ - 20mmHg DBP St - Su $\le$ - 10mmHg Su SBP $\ge$ 160 mmHg - SBP St - Su $\le$ - 30 mmHg DBP St - Su $\le$ - 15 mmHg Orthostatic PR $\ge$ 30 beats/min | |
| Weight | >5% increase from baseline<br>>5% decrease from baseline | FDA Feb 2007. |


Mitsubishi Tanabe Pharma Corporation

| Parameter | PCSV | Comments |
|---|---|---|
| ECG: Ref.: | ECG: Ref.: CPMP 1997 guideline. ICH E14 2005 | |
| HR | ≤50 bpm and decrease from baseline≥20 bpm | |
| | >120 bpm and increase from baseline<br>>20 bpm | |
| PR | >220 ms and increase from baseline | |
| QRS | $\geq$ 120 ms & < 120 ms at baseline | |
| QTc | Absolute values (ms) | To be applied to QTcF formula. |
| | >450 ms and baseline <=450 ms<br>>480 ms and baseline <=480 ms<br>>500 ms and <=500 ms at baseline | |
| | Increase from baseline 30-60 ms<br>Increase from baseline >60 ms | |
| | | : |

**Appendix 3** Reference Value in Each Laboratory Parameters

| Parameter | Reference Value |
|----------------------------|--------------------------------|
| RBC count (10^12/L) | Male |
| | Low $< 4.3$ , High $> 5.7$ |
| | Female |
| | Low < 3.8, High > 5 |
| Hemoglobin (g/L) | Male |
| | Low < 135, High > 175 |
| | Female |
| | Low < 115, High > 150 |
| Hematocrit (L/L) | Male |
| | Low $< 0.397$ , High $> 0.524$ |
| | Female |
| · . | Low < 0.348, High > 0.45 |
| MCHC (g/dL) | Low < 30.2, High > 35.1 |
| WBC count (10^9/L) | Low < 3.3, High > 9 |
| Platelet count (10^9/L) | Low < 140, High > 340 |
| AST (GOT) (U/L) | Low < 10, High > 40 |
| ALT (GPT) (U/L) | Low < 5, High > 45 |
| ALP (U/L) | Low < 100, High > 325 |
| LDH (U/L) | Low < 120, High > 240 |
| Gamma-GTP (U/L) | Male |
| | High > 80 |
| | Female |
| | High > 30 |
| Total protein (g/L) | Low < 67, High > 83 |
| Albumin (g/L) | Low < 38, High > 52 |
| Total cholesterol (mmol/L) | Low < 3.108, High > 5.672 |
| Total bilirubin (umol/L) | Low < 3.421, High > 20.525 |
| BUN (mmol/L) | Low < 2.856, High > 7.14 |
| Serum creatinine (umol/L) | Male |
| | Low < 53.925, High > 91.938 |
| | Female |
| | Low < 41.549, High > 69.838 |

| Parameter | Reference Value |
|-------------------------------|-------------------------------|
| Na (mmol/L) | Low < 137, High > 147 |
| K (mmol/L) | Low < 3.5, High > 5 |
| Cl (mmol/L) | Low < 98, High > 108 |
| Ca (mmol/L) | Low < 2.1, High > 2.6 |
| HCO3- (mmol/L) | Low < 19.2, High > 27.1 |
| Uric acid (umol/L) | Male |
| | Low < 226.043, High > 416.395 |
| | Female |
| | Low < 148.713, High > 416.395 |
| Triglycerides (mmol/L) | Low < 0.339, High > 1.684 |
| BAP (ug/L) | Male |
| | Low $< 3.7$ , High $> 20.9$ |
| | Female |
| | Premenopause(30 - 44 years) |
| | Low $< 2.9$ , High $> 14.5$ |
| | Postmenopausal(45 - 79 years) |
| | Low $< 3.8$ , High $> 22.6$ |
| Inorganic phosphorus (mmol/L) | Low < 0.808, High > 1.454 |
| CPK (U/L) | Male |
| | Low $< 40$ , High $> 150$ |
| | Female |
| | Low < 60, High > 270 |
| CRP (mg/L) | High > 3 |





# APPROVAL FORM

# Statistical Analysis Plan(For Database at Week 68)

|---|---|
| Protocol Title | A Phase 2/3 (Placebo-Controlled, Double-Blind, Comparative) Study<br>on MT-5547 in Patients with Osteoarthritis Accompanied by<br>Moderate to Severe Pain |
| Version / Date | 1.0 / 19-April-2021 |

### Authors:

| Statistics Author | |
|--------------------|------------------|
| Print Name: | |
| Position: | Biostatistician |
| Clinical Pharmacol | kinetica Author |
| Print Name: | |
| Position: | Pharmacokinetics |

#### Approved by:

| Statistic Approver | k je <u>livideratife kie, i er er er er</u> |
|--------------------|---------------------------------------------|
| Print Name: | |
| Position: | Responsible Biostatistician |
| Signature: | Refer to email |
| Approval date: | Refer to email |
| Clinical Pharmaco | kinetic Approver |
| Print Name: | |
| Position: | Responsible Pharmacokinetics |
| Signature: | Refer to email |
| Approval date: | Refer to email |




# APPROVAL FORM

# Statistical Analysis Plan(For Database at Week 68)

| Protocol No. | MT-5547-301 |
|---|---|
| Protocol Tale | A Phase 2/3 (Placebo-Controlled, Double-Bland, Comparative) Study |
| | on MT-5547 in Patients with Osteoarthritis Accompanied by |
| | Moderate to Severe Pain |
| Version Date | 1.0 · 19-April-2021 |

| Statistics Author | Transfer Section 1 |
|--------------------|--------------------|
| Print Name: | |
| Position: | Biostatistician |
| Clinical Pharmacol | cinetics Author |
| Print Name: | |
| Position: | Pharmacokinetics |

| Statistic Approver | |
|--------------------|------------------------------|
| Print Name: | |
| Position: | Responsible Biostatistician |
| Signature: | Refer to email |
| Approval date: | Refer to email |
| Clinical Pharmaco | kinetic Approver |
| Print Name: | |
| Positios: | Responsible Pharmacokinetics |
| Signature: | Refer to email |
| Approval date: | Refer to email |


colidectal